CLINICAL TRIAL: NCT02699736
Title: EuroSIDA Prospective Observational Cohort Study on Clinical and Virological Outcome of European Patients Infected With HIV
Brief Title: EuroSIDA - Clinical and Virological Outcome of European Patients Infected With HIV
Acronym: EuroSIDA
Status: Enrolling by invitation | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Jens D Lundgren, MD, CHIP Administrative Director, Rigshospitalet, Denmark
Other Study IDs: The EuroSIDA Study; QLK2-2000-00773 (Other Grant/Funding Number: EC FP5 1998-2002); LSHC-CT-2006-018632 (Other Grant/Funding Number: EC FP6 2002-2006); Gilead EuroSIDA (Other Grant/Funding Number: Gilead); GSK EuroSIDA (Other Grant/Funding Number: GlaxoSmithKline); Janssen EuroSIDA (Other Grant/Funding Number: Janssen); CT94-1637 (Other Grant/Funding Number: EC BIOMED 1); CT97-2713 (Other Grant/Funding Number: EC BIOMED 2); Pfizer EuroSIDA (Other Grant/Funding Number: Pfizer); Merck EuroSIDA (Other Grant/Funding Number: Merck and Co); BMS EuroSIDA (Other Grant/Funding Number: Bristol-Myers Squibb); SNSF 108787 (Other Grant/Funding Number: The Swiss National Science Foundation)
Record Dates: First submitted 2016-01-19; First posted 2016-03-04 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: HIV; Hepatitis B; Hepatitis C; AIDS; Coinfection; Cardiovascular Diseases; Diabetes Mellitus; Acidosis, Lactic; Renal Insufficiency; Fractures, Bone; End Stage Liver Disease; Kidney Failure, Chronic; Proteinuria
Keywords: HIV; HIV-1; Hepatitis C; HCV; prospective; cohort; coinfection
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Acquired Immunodeficiency Syndrome; Coinfection; Cardiovascular Diseases; Diabetes Mellitus; Acidosis, Lactic; Renal Insufficiency; Fractures, Bone; End Stage Liver Disease; Kidney Failure, Chronic; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples Without DNA — 2 x 1 ml plasma;
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (11):
- Cohort I: Enrolled from August 1994. Patients to be included were those attending the out-patient clinic for a scheduled visit (i.e. appointment made more than 2 weeks before time of visit). For patients included in the study from 1994-1997, it was requested that the patients had a cluster of differentiation 4 (CD4) count < 500 cells/µL within the last 5 months before inclusion. For all HIV patients enrolled and under follow up, laboratory, therapeutic and clinical data are collected twice annually. Demographic data, date on pregnancy and serological evidence for infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.
- Cohort II: Enrolled from January 1996. Patients to be included were those attending the out-patient clinic for a scheduled visit (i.e. appointment made more than 2 weeks before time of visit). For patients included in the study from 1994-1997, it was requested that the patients had a cluster of differentiation 4 (CD4) count < 500 cells/µL within the last 5 months before inclusion. For all HIV patients enrolled and under follow up, laboratory, therapeutic and clinical data are collected twice annually. Demographic data, date on pregnancy and serological evidence for infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.
- Cohort III: Enrolled from February 1997. Patients to be included were those attending the out-patient clinic for a scheduled visit (i.e. appointment made more than 2 weeks before time of visit). For patients included in the study from 1994-1997, it was requested that the patients had a cluster of differentiation 4 (CD4) count < 500 cells/µL within the last 5 months before inclusion. For all HIV patients enrolled and under follow up, laboratory, therapeutic and clinical data are collected twice annually. Demographic data, date on pregnancy and serological evidence for infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.
- Cohort IV: Enrolled from March 1999. Patients to be included were those attending the out-patient clinic for a scheduled visit (i.e. appointment made more than 2 weeks before time of visit). The eligibility criteria of a cluster of differentiation 4 (CD4) count < 500 cells/µL within the last 5 months before inclusion has been removed for patients joining the study in 1999 and beyond, since the intention of the study is to include most patients eligible for antiretroviral therapy. For all HIV patients enrolled and under follow up, laboratory, therapeutic and clinical data are collected twice annually. Demographic data, date on pregnancy and serological evidence for infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.
- Cohort V: Patients to be included were those aged 16 years or older attending the out-patient clinic for a scheduled visit (i.e. appointment made more than 2 weeks before time of visit), regardless of cluster of differentiation 4 (CD4) cell count. For all HIV patients enrolled and under follow up, laboratory, therapeutic and clinical data are collected twice annually. Demographic data, date on pregnancy and serological evidence for infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.
- Cohort VI: Patients to be included were those aged 16 years or older attending the out-patient clinic for a scheduled visit (i.e. appointment made more than 2 weeks before time of visit), regardless of cluster of differentiation 4 (CD4) cell count. For all HIV patients enrolled and under follow up, laboratory, therapeutic and clinical data are collected twice annually. Demographic data, date on pregnancy and serological evidence for infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.
- Cohort VII: Patients to be included were those aged 16 years or older attending the out-patient clinic for a scheduled visit (i.e. appointment made more than 2 weeks before time of visit), regardless of cluster of differentiation 4 (CD4) cell count. For all HIV patients enrolled and under follow up, laboratory, therapeutic and clinical data are collected twice annually. Demographic data, date on pregnancy and serological evidence for infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.
- Cohort VIII: Patients to be included were those aged 16 years or older attending the out-patient clinic for a scheduled visit (i.e. appointment made more than 2 weeks before time of visit), regardless of cluster of differentiation 4 (CD4) cell count. For all HIV patients enrolled and under follow up, laboratory, therapeutic and clinical data are collected twice annually. Demographic data, date on pregnancy and serological evidence for infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.
- Cohort IX: Enrolled from December 2011. Patients to be included were those aged 16 years or older attending the out-patient clinic for a scheduled visit (i.e. appointment made more than 2 weeks before time of visit), regardless of cluster of differentiation 4 (CD4) cell count. For all HIV patients enrolled and under follow up, laboratory, therapeutic and clinical data are collected twice annually. Demographic data, date on pregnancy and serological evidence for infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.
- Cohort X: All patients should be consecutive patients (except those already enrolled in EuroSIDA), or patients who had a scheduled visit (i.e. those who made an appointment >2 weeks prior to their visit) in the outpatient clinic regardless of cluster of differentiation 4 (CD4) cell count and ART status). Enroll patients of 16 years or older and positive for antibodies against hepatitis C virus (regardless of HCV-RNA status, fibrosis stage and prior treatment against hepatitis C). For all HIV patients enrolled and under follow up, laboratory, therapeutic and clinical data are collected twice annually. Demographic data, date on pregnancy and serological evidence for infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.
- Cohort XI: HIV-1 positive persons ≥18 years of age, not already enrolled in EuroSIDA, are eligible for inclusion. Participants should be enrolled consecutively in one of the following two groups:
  1. Participants who have started integrase inhibitor (INSTI) based antiretroviral therapy (ART) after 1/1/2012 and have a CD4 cell count and HIV-RNA available in the 12 months prior to starting INSTI or within 3 months after starting INSTI
  2. If participants have not started INSTI, they should be included providing they have a CD4/HIV-RNA in the 12 months prior to baseline or within 3 months after baseline.
  For all patients enrolled and under follow up, laboratory, therapeutic, clinical and demographic data, date on pregnancy and data on hepatitis B virus (HBV) and hepatitis C virus (HCV) are collected once annually.

SUMMARY:
The EuroSIDA study is a prospective observational cohort study of 23,000+ patients followed in 100+ clinics in 35 European countries, Israel and Argentina. The study is the largest pan-European cohort study and few studies of a comparable design are available on a global scale. The EuroSIDA study is an ongoing collaboration and patients have been enrolled into the study through 11 cohorts since 1994.

The main objective of the study remains the same as in 1994: to prospectively study, clinical, therapeutic, demographic, virological and laboratory data from HIV-1 positive persons across Europe in order to determine their long-term virological, immunological and clinical outcomes.

Historically, EuroSIDA has been crucial in reporting key changes in the HIV epidemic, such as the dramatic changes in morbidity and mortality when combination anti-retroviral therapy (cART) was first introduced. As new anti-HCV treatment is introduced to HIV/HCV co-infected patients, it is important for EuroSIDA to remain in the forefront of investigating the treatment benefits and adverse effects.

All study documents, study status, newsletters, scientific publications and presentations are available online and are updated continuously at project website.

In general terms, the objective of the EuroSIDA study is to continue a long-term, prospective collection of clinical, laboratory and therapeutic data as well as plasma on a large cohort of consecutive HIV infected patients from across Europe in order to (1) assess the factors associated with the clinical, immunological and virological course of HIV infection and HIV-related co-infections and co-morbidities, and (2) continue to provide and develop a surveillance system to describe temporal changes and regional differences in the clinical course of HIV and HIV-related co-infections and co-morbidities in Europe.

DETAILED DESCRIPTION:
Abstract: There are currently over 1½ million people across Europe infected with HIV. The epidemic continues to intensify in the Eastern European region where prevalence of HIV will continue to increase in the years to come. There are significant problems with the management of this public health crisis. Available antiretroviral therapy (ART) - although extremely effective - does not eradicate HIV and hence has to be continued for life. Other limitations are the development of resistance, adverse effects of treatment, and the requirement for strict adherence. Despite these limitations, the widespread use of potent ART has resulted in a dramatic decrease in HIV-related mortality across Europe. As the incidence of AIDS has declined, the relative importance of co-morbidities and co-infections, such as chronic viral hepatitis and tuberculosis (TB), has increased. Around a third of all EuroSIDA patients are co-infected with hepatitis C virus (HCV), and liver-related death is now the second most common cause of death after AIDS. With the introduction of new more potent and better tolerated oral direct acting antivirals (DAAs) against HCV, major changes in the management and outcome HCV co-infection is anticipated in the coming years. However due to the high cost of DAAs, access to new treatment could vary substantially across Europe.

Over 23,000 consecutively enrolled HIV-1 positive patients from over 100 clinical centres in 35 European countries, Israel and Argentina - one quarter from the eastern region - are currently enrolled in EuroSIDA. New cohorts of patients are normally enrolled every 2-3 years to ensure all regions of Europe where the epidemic is prevalent are represented so the study will give timely information on the clinical presentation and outcome of European HIV-1 positive patients. In 2012, 2500 additional patients were enrolled into EuroSIDA cohort IX. To be at the forefront of investigating the benefits and adverse effects of new HCV treatment in co-infected patients, the EuroSIDA cohort X enrolled in 2014, consisted of 4000 HIV-1 patients positive for antibodies against HCV. The next cohort to be enrolled (cohort XI) in 2019 will consist of 1500 HIV-1 positive patients.

The EuroSIDA study group has now been working on the EuroSIDA study since 1994 and has several notable accomplishments to date, including publication of more than 200 papers in peer-reviewed journals (including the New England Journal of Medicine and the Lancet among others). The focus of EuroSIDA has naturally changed over this period, which demonstrates an eagerness to be flexible, dynamic, and focus on contemporary issues, and the study group is committed to continue working with such principles.

In recent years, EuroSIDA has, in addition to the scientific publications, prioritized capacity building in Eastern Europe with HIV seminars, hosting clinicians from Eastern Europe as European AIDS Clinical Society (EACS) students in the office of Copenhagen HIV Programme and sponsoring 2-3 young physicians from Eastern Europe to participate in a statistical course in London every year.

Most of the data are collected from the clinics as part of routine care. Additionally, the central plasma repository will be used to extend earlier studies of the viral epidemiology of HIV (resistance and subtypes).

Primary study objective: To prospectively study, clinical, therapeutic, demographic, virological and laboratory data from HIV-1 positive persons across Europe in order to determine the long-term virological, immunological and clinical outcome. The specific objectives, falling into four main categories, are as follows:

1. To examine the efficacy of ART and factors that limits this
2. To detect current or emerging late onset adverse events among patients on ART
3. To continue surveillance of HIV in clinics around Europe to describe temporal changes and regional difference
4. To monitor the uptake and outcome of HCV therapy and development of direct acting antivirals and compare differences between EuroSIDA regions

Study visits: Enrolment + follow-up Data collection: For all HIV-1 positive patients enrolled and under follow up, laboratory, therapeutic and clinical data on HIV, viral hepatitis and serious non-AIDS clinical events are collected, as well as demographic data and possible data on pregnancy and the HIV status of the newborn baby. The patients are seen within their clinics as required and according to their local physician. EuroSIDA does not involve patient interviews or study visits, the information is collected from patient notes twice a year until 2017 hereafter once a year.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients regardless of CD4 cell count and ART status
* Must be positive for antibodies against HCV regardless of HCV-RNA status, fibrosis stage and prior HCV therapy

Exclusion Criteria:

* Patients under 16 years of age
* Already enrolled in EuroSIDA through earlier cohort
* Predefined number of patients has been reached

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The EuroSIDA study recruits HIV-1 positive patients above the age of 16 years in the proportions in which they are represented in the participating clinics, which ensures that women are proportionally represented in the study. Approximately 26% of the patients are women. The study does not intervene with the clinical management of the patients followed, but only collects information based on provider-patient interviews, from patient records and from plasma samples collected. Pregnant women may participate in the study, as no interference with their treatment or pregnancy in any way will take place. Data on frequency and outcome of pregnancy are collected in the study once a year.
Sampling Method: Non-Probability Sample
Enrollment: 23000 (Estimated)
Dates: Start 1994-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of long-term virological, immunological and morbidity and mortality outcomes across different regions in Europe; and demographic, clinical, therapeutic and viral factors associated with these outcomes | From date of enrollment until the date of progression, lost to follow-up or death, whichever came first, assessed up to 5 years
  EuroSIDA is a non-interventional epidemiological cohort study that collects structured data. Data is not collected real time, but in 6-monthly intervals. The clinical data is centered on collecting laboratory variables and ascertaining predefined meaningful clinical events as well as reasons for changing and or stopping treatment regimens. The observational cohort study concept means that EuroSIDA does not collect Adverse Events, Adverse Reactions, Serious Adverse Reactions or Suspected Unexpected Serious Adverse Reactions as defined by pharmacovigilance requirements for marketing authorization holders. However, EuroSIDA often analyses and reports specific clinical events of interest, occasionally related to drug classes, but more regularly with a focus on regional differences in treatment and care.

SECONDARY OUTCOMES:
Number of patients experiencing HIV-related events over time | From date of enrollment until the date of progression, lost to follow-up or death, whichever came first, assessed up to 5 years
Number of participants experiencing HIV-related events by region | From date of enrollment until the date of progression, lost to follow-up or death, whichever came first, assessed up to 5 years
Proportion of HCV infected patients who start treatment with direct acting antiretrovirals | From date of enrollment until the date of progression, lost to follow-up or death, whichever came first, assessed up to 5 years
Rate of sustained virologic response 12 (SVR12) in HCV-infected patients | From date of enrollment until the date of progression, lost to follow-up or death, whichever came first, assessed up to 5 years
  Share of patients with undetectable viral load 12 weeks after cessation of therapy targeting HCV infection
Incidence of liver-related clinical outcomes in HCV-infected patients receiving HCV therapy | From date of enrollment until the date of progression, lost to follow-up or death, whichever came first, assessed up to 5 years
Incidence of non-liver-related clinical outcomes in HCV-infected patients receiving HCV therapy | From date of enrollment until the date of progression, lost to follow-up or death, whichever came first, assessed up to 5 years
Incidence of liver-related clinical outcomes in HCV-infected patients not receiving HCV therapy | From date of enrollment until the date of progression, lost to follow-up or death, whichever came first, assessed up to 5 years
Incidence of non-liver-related clinical outcomes in HCV-infected patients not receiving HCV therapy | From date of enrollment until the date of progression, lost to follow-up or death, whichever came first, assessed up to 5 years
Incidence of toxicities related to direct acting antivirals by regions | From date of enrollment until the date of progression, lost to follow-up or death, whichever came first, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Wandeler, Dr. med., Study Chair — University of Bern, Switzerland.
Locations (110):
- Hospital JM Ramos Mejia, Buenos Aires, Argentina
- Austria (2):
  - Medical University Insbruck, Innsbruck
  - Otto Wagner Spital, Vienna
- Belarus (3):
  - GOCGEIOZ - Gomel Regional Centre for Hygiene, Homyel
  - Gomel State Medical University, Homyel
  - Belarus State Medical University, Minsk
- Belgium (3):
  - Institute of Tropical Medicine, Antwerp
  - CHU Saint-Pierre, Brussels
  - University Ziekenhuis Gent, Ghent
- Klinicki centar Univerziteta Sarajevo (KCUS), Sarajevo, Bosnia and Herzegovina
- University Hospital of Infectious Diseases, Zagreb, Croatia
- Czechia (2):
  - Charles University Hospital Plzeň, Pilsen
  - Faculty Hospital Bulovka, Prague
- Denmark (6):
  - Rigshospitalet, Copenhagen
  - Hilleroed Sygehus, Hillerød
  - Hvidovre Universitets Hospital, Hvidovre
  - Odense Universitetshospital, Odense
  - Roskilde Sygehus, Roskilde
  - Aarhus Universitetshospital Skejby, Skejby
- Estonia (2):
  - Narva AIDS Centre, Kohtla-Järve
  - West-Tallinn Central Hospital, Tallinn
- Helsinki University Central Hospital, Helsinki, Finland
- France (8):
  - INSERM, Université Bordeaux Segalen, Bordeaux
  - Hopital Edouard Herriot, Lyon
  - Hospital de la Croix Rousse, Lyon
  - CHU Nice Hopital de l' Archet 1, Nice
  - Hospital Saint Antoine, Paris
  - Hôpital de la Pitié-Salpétière, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôtel-Dieu Hospital, Paris
- Georgian AIDS and Clinical Immunology Research Center, Tbilisi, Georgia
- Germany (8):
  - University Hospital Bonn, Bonn
  - University Hospital Cologne, Cologne
  - University Clinic Hamburg Eppendorf, Eppendorf
  - J.W.Goethe University Hospital, Frankfurt am Main
  - Bernhard Nocht Institut für Tropenmedizin, Hamburg
  - ICH Study Center, Hamburg
  - Mediziniche Hochschule Hannover, Hanover
  - Ludwig-Maximilians-Universität, Medizinische Poliklinik, München
- Greece (3):
  - 1st I.K.A Hospital of Athens, Athens
  - Ippokration General Hospital, Athens
  - The General Hospital of Athens "G. Gennimatas", Athens
- Szent László Hospital, Budapest, Hungary
- Landspitali University Hospital, Reykjavik, Iceland
- St. James' Hospital, Dublin, Ireland
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah Hospital, Jerusalem
  - Kaplan Medical Center, AIDS Center Neve Or, Rehovot
  - Ichilov Hospital, Tel Aviv
- Italy (8):
  - Ospedale Riuniti, Divisione Malattie Infettive, Bergamo
  - Ospedale L. Sacco, Milan
  - Ospedale San Paulo, Milan
  - Ospedale San Raffaele, Milan
  - Università degli Studi di Modena, Modena
  - Ospedale Cotugno, III Divisione Malattie Infettive, Napoli
  - National Institute for Infectious Diseases, Rome
  - Poloclinico Umberto 1, Rome
- Infectology Center of Latvia, Riga, Latvia
- Lithuania (2):
  - Infectious Diseases and Tuberculosis Hospital, Vilnius University Hospital branch, Vilnius
  - Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Academisch Ziekenhuis bij de Universiteit van Amsterdam, Amsterdam, Netherlands
- Oslo Universitetssykehus, Oslo, Norway
- Poland (8):
  - Uniwersytecki Szpital Kliniczny, Bialystok
  - Szpital Specjalistyczny, Osrodek Diagnostyki i Terapii AIDS, Chorzów
  - Medical University Gdansk, Gdansk
  - Wojewodzki Szpital Specjalistyczny im. WI. Bieganskiego, Lodz
  - Poznan University of Medical Sciences, Poznan
  - Pomeramian Academy of Medicine (PAM), Szczecin
  - Wojewodzki Szpital Zakazny, Warsaw
  - EMC Instytut Medyczny SA, Wroclaw
- Portugal (3):
  - Hospital Curry Cabral, Lisbon
  - Hospital de Egas Moniz, Lisbon
  - Hospital Santa Maria, Lisbon
- Dr. Victor Babes Hospital, Bucharest, Romania
- Russia (4):
  - Centre for HIV/AIDS & and infectious diseases, Kaliningrad
  - Nizhny Novgorod Scientific and Research Institute, Nizhny Novgorod
  - St Petersburgs AIDS Centre, Saint Petersburg
  - Novgorod Centre for AIDS prevention and control, Veliky Novgorod
- The Institute for Infectious and Tropical Diseases, Belgrade, Serbia
- Slovak Medical University, Bratislava, Slovakia
- University Clinical Centre Ljubljana, Ljubljana, Slovenia
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clínic, University of Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Carlos III, Departamento de Enfermedades Infecciosas, Madrid
  - Hospital La Paz, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Consorcio Hospital General Universitario Valencia, Valencia
  - Hospital Universitario de Alava, Vitoria-Gasteiz
- Sweden (3):
  - Skåne University Hospital, Malmo
  - Karolinska University Hospital Huddinge, Stockholm
  - Södersjukhuset, Stockholm
- Switzerland (6):
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern
  - Hopital Cantonal Universitaire Geneve, Geneva
  - Centre hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - University Hospital Zürich, Zurich
- Ukraine (5):
  - Kharkiv State Medical University, Kharkiv
  - Luhansk AIDS Center, Luhansk
  - Lviv Regional HIV/AIDS Prevention and Control CTR, Lviv
  - Odessa Region AIDS Center, Odesa
  - Crimean Republican AIDS centre, Simferopol
- United Kingdom (6):
  - Royal Sussex County Hospital, Brighton
  - Western General Hospital, Edinburgh
  - Royal London Hospital, London
  - St. Mary's Hospital, London
  - University College London, Mortimer Market Centre, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill A, Grossman H, Cohen C, Nadler J, Peeters M. Modelling-based prediction of clinical benefits from etravirine in the TMC125-C223 trial. HIV Clin Trials. 2007 Mar-Apr;8(2):68-76. doi: 10.1310/hct0802-68. PMID 17507322
- [Background] Carter M. EuroSIDA cohort: 9% coinfected with HIV/HBV. IAPAC Mon. 2005 Apr;11(4):110. No abstract available. PMID 16110550
- [Result] Podlekareva D, Grint D, Karpov I, Rakmanova A, Mansinho K, Chentsova N, Zeltina I, Losso M, Parczewski M, Lundgren JD, Mocroft A, Kirk O; EuroSIDA in EuroCoord. Changing utilization of Stavudine (d4T) in HIV-positive people in 2006-2013 in the EuroSIDA study. HIV Med. 2015 Oct;16(9):533-43. doi: 10.1111/hiv.12254. Epub 2015 May 18. PMID 25988795
- [Result] Shepherd L, Borges AH, Ravn L, Harvey R, Jean-Paul V, Bower M, Grulich A, Silverberg M, De Wit S, Kirk O, Lundgren J, Mocroft A; EuroSIDA in Eurocoord. Predictive value of prostate-specific antigen for prostate cancer: a nested case-control study in EuroSIDA. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19510. doi: 10.7448/IAS.17.4.19510. eCollection 2014. PMID 25394019
- [Result] Laut KG, Mocroft A, Lazarus J, Reiss P, Rockstroh J, Karpov I, Rakhmanova A, Knysz B, Moreno S, Gargalianos P, Lundgren J, Kirk O; Eurosida in Eurocoord. Regional differences in self-reported HIV care and management in the EuroSIDA study. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19504. doi: 10.7448/IAS.17.4.19504. eCollection 2014. PMID 25394013
- [Result] Peters L, Mocroft A, Lundgren J, Grint D, Kirk O, Rockstroh J. HIV and hepatitis C co-infection in Europe, Israel and Argentina: a EuroSIDA perspective. BMC Infect Dis. 2014;14 Suppl 6(Suppl 6):S13. doi: 10.1186/1471-2334-14-S6-S13. Epub 2014 Sep 19. No abstract available. PMID 25253564
- [Result] Grint D, Peters L, Schwarze-Zander C, Beniowski M, Pradier C, Battegay M, Jevtovic D, Soriano V, Lundgren JD, Rockstroh JK, Kirk O, Mocroft A; EuroSIDA in EuroCoord. Temporal changes and regional differences in treatment uptake of hepatitis C therapy in EuroSIDA. HIV Med. 2013 Nov;14(10):614-23. doi: 10.1111/hiv.12068. Epub 2013 Jul 19. PMID 23869664
- [Result] Podlekareva DN, Reekie J, Mocroft A, Losso M, Rakhmanova AG, Bakowska E, Karpov IA, Lazarus JV, Gatell J, Lundgren JD, Kirk O; EuroSIDA study in EuroCoord. Benchmarking HIV health care: from individual patient care to health care evaluation. An example from the EuroSIDA study. BMC Infect Dis. 2012 Sep 25;12:229. doi: 10.1186/1471-2334-12-229. PMID 23009317
- [Result] Reekie J, Kowalska JD, Karpov I, Rockstroh J, Karlsson A, Rakhmanova A, Horban A, Kirk O, Lundgren JD, Mocroft A; EuroSIDA in EuroCoord. Regional differences in AIDS and non-AIDS related mortality in HIV-positive individuals across Europe and Argentina: the EuroSIDA study. PLoS One. 2012;7(7):e41673. doi: 10.1371/journal.pone.0041673. Epub 2012 Jul 23. PMID 22911841
- [Result] Fox ZV, Cozzi-Lepri A, D'Arminio Monforte A, Karlsson A, Phillips AN, Kronborg G, Kjaer J, Clotet B, Lundgren JD; EuroSIDA. Predictors of having a resistance test following confirmed virological failure of combination antiretroviral therapy: data from EuroSIDA. Antivir Ther. 2011;16(5):781-5. doi: 10.3851/IMP1801. PMID 21817201
- [Result] Viard JP, Souberbielle JC, Kirk O, Reekie J, Knysz B, Losso M, Gatell J, Pedersen C, Bogner JR, Lundgren JD, Mocroft A; EuroSIDA Study Group. Vitamin D and clinical disease progression in HIV infection: results from the EuroSIDA study. AIDS. 2011 Jun 19;25(10):1305-15. doi: 10.1097/QAD.0b013e328347f6f7. PMID 21522006
- [Result] Kowalska JD, Mocroft A, Ledergerber B, Florence E, Ristola M, Begovac J, Sambatakou H, Pedersen C, Lundgren JD, Kirk O; Eurosida Study Group. A standardized algorithm for determining the underlying cause of death in HIV infection as AIDS or non-AIDS related: results from the EuroSIDA study. HIV Clin Trials. 2011 Mar-Apr;12(2):109-17. doi: 10.1310/hct1202-109. PMID 21498154
- [Result] Reekie J, Reiss P, Ledergerber B, Sedlacek D, Parczewski M, Gatell J, Katlama C, Fatkenheuer G, Lundgren JD, Mocroft A; EuroSIDA study group. A comparison of the long-term durability of nevirapine, efavirenz and lopinavir in routine clinical practice in Europe: a EuroSIDA study. HIV Med. 2011 May;12(5):259-68. doi: 10.1111/j.1468-1293.2010.00877.x. Epub 2010 Aug 31. PMID 20812948
- [Result] van Luin M, Bannister WP, Mocroft A, Reiss P, Di Perri G, Peytavin G, Molto J, Karlson A, Castagna A, Beniowski M, Lundgren JD, Burger DM; EuroSIDA Study Group. Absence of a relation between efavirenz plasma concentrations and toxicity-driven efavirenz discontinuations in the EuroSIDA study. Antivir Ther. 2009;14(1):75-83. PMID 19320239
- [Result] Podlekareva D, Bannister W, Mocroft A, Abrosimova L, Karpov I, Lundgren JD, Kirk O; EuroSIDA Study Group. The EuroSIDA study: Regional differences in the HIV-1 epidemic and treatment response to antiretroviral therapy among HIV-infected patients across Europe--a review of published results. Cent Eur J Public Health. 2008 Sep;16(3):99-105. doi: 10.21101/cejph.a3490. PMID 18935770
- [Result] Bannister WP, Friis-Moller N, Mocroft A, Viard JP, van Lunzen J, Kirk O, Gargalianos P, Banhegyi D, Chiesi A, Lundgren JD; EuroSIDA Study Group. Incidence of abacavir hypersensitivity reactions in euroSIDA. Antivir Ther. 2008;13(5):687-96. PMID 18771052
- [Result] Bannister WP, Cozzi-Lepri A, Clotet B, Mocroft A, Kjaer J, Reiss P, von Wyl V, Lazzarin A, Katlama C, Phillips AN, Ruiz L, Lundgren JD; EuroSIDA study group. Transmitted drug resistant HIV-1 and association with virologic and CD4 cell count response to combination antiretroviral therapy in the EuroSIDA Study. J Acquir Immune Defic Syndr. 2008 Jul 1;48(3):324-33. doi: 10.1097/QAI.0b013e31817ae5c0. PMID 18545152
- [Result] Bannister WP, Ruiz L, Cozzi-Lepri A, Mocroft A, Kirk O, Staszewski S, Loveday C, Karlsson A, Monforte Ad, Clotet B, Lundgren JD; EuroSIDA study group. Comparison of genotypic resistance profiles and virological response between patients starting nevirapine and efavirenz in EuroSIDA. AIDS. 2008 Jan 30;22(3):367-76. doi: 10.1097/QAD.0b013e3282f3cc35. PMID 18195563
- [Result] Fessel J, Hurley LB. Incidence of pancreatitis in HIV-infected patients: comment on findings in EuroSIDA cohort. AIDS. 2008 Jan 2;22(1):145-7. doi: 10.1097/QAD.0b013e3282f030a9. No abstract available. PMID 18090403
- [Result] Smith CJ, Olsen CH, Mocroft A, Viard JP, Staszewski S, Panos G, Staub T, Blaxhult A, Vetter N, Lundgren JD. The role of antiretroviral therapy in the incidence of pancreatitis in HIV-positive individuals in the EuroSIDA study. AIDS. 2008 Jan 2;22(1):47-56. doi: 10.1097/QAD.0b013e3282f03094. PMID 18090391
- [Result] Mocroft A, Ledergerber B, Zilmer K, Kirk O, Hirschel B, Viard JP, Reiss P, Francioli P, Lazzarin A, Machala L, Phillips AN, Lundgren JD; EuroSIDA study group and the Swiss HIV Cohort Study. Short-term clinical disease progression in HIV-1-positive patients taking combination antiretroviral therapy: the EuroSIDA risk-score. AIDS. 2007 Sep 12;21(14):1867-75. doi: 10.1097/QAD.0b013e328270b877. PMID 17721094
- [Result] Podlekareva D, Mocroft A, Dragsted UB, Ledergerber B, Beniowski M, Lazzarin A, Weber J, Clumeck N, Vetter N, Phillips A, Lundgren JD; EuroSIDA study group. Factors associated with the development of opportunistic infections in HIV-1-infected adults with high CD4+ cell counts: a EuroSIDA study. J Infect Dis. 2006 Sep 1;194(5):633-41. doi: 10.1086/506366. Epub 2006 Jul 24. PMID 16897662
- [Result] Konopnicki D, Mocroft A, de Wit S, Antunes F, Ledergerber B, Katlama C, Zilmer K, Vella S, Kirk O, Lundgren JD; EuroSIDA Group. Hepatitis B and HIV: prevalence, AIDS progression, response to highly active antiretroviral therapy and increased mortality in the EuroSIDA cohort. AIDS. 2005 Mar 24;19(6):593-601. doi: 10.1097/01.aids.0000163936.99401.fe. PMID 15802978
- [Result] Mocroft A, Monforte Ad, Kirk O, Johnson MA, Friis-Moller N, Banhegyi D, Blaxhult A, Mulcahy F, Gatell JM, Lundgren JD; EuroSIDA study group. Changes in hospital admissions across Europe: 1995-2003. Results from the EuroSIDA study. HIV Med. 2004 Nov;5(6):437-47. doi: 10.1111/j.1468-1293.2004.00250.x. PMID 15544697
- [Result] Cabrera C, Cozzi-Lepri A, Phillips AN, Loveday C, Kirk O, Ait-Khaled M, Reiss P, Kjaer J, Ledergerber B, Lundgren JD, Clotet B, Ruiz L; EuroSIDA Study Group. Baseline resistance and virological outcome in patients with virological failure who start a regimen containing abacavir: EuroSIDA study. Antivir Ther. 2004 Oct;9(5):787-800. PMID 15535417
- [Result] Mocroft A, Ledergerber B, Viard JP, Staszewski S, Murphy M, Chiesi A, Horban A, Hansen AB, Phillips AN, Lundgren JD; EuroSIDA Study Group. Time to virological failure of 3 classes of antiretrovirals after initiation of highly active antiretroviral therapy: results from the EuroSIDA study group. J Infect Dis. 2004 Dec 1;190(11):1947-56. doi: 10.1086/425424. Epub 2004 Oct 28. PMID 15529259
- [Result] Kirk O, Mocroft A, Lundgren JD; EuroSIDA-studiet. [Decline in AIDS and death rates in the EuroSIDA study. An observational study]. Ugeskr Laeger. 2004 Jun 21;166(26-31):2572-6. No abstract available. Danish. PMID 15285167
- [Result] Yust I, Fox Z, Burke M, Johnson A, Turner D, Mocroft A, Katlama C, Ledergerber B, Reiss P, Kirk O; EuroSIDA. Retinal and extraocular cytomegalovirus end-organ disease in HIV-infected patients in Europe: a EuroSIDA study, 1994-2001. Eur J Clin Microbiol Infect Dis. 2004 Jul;23(7):550-9. doi: 10.1007/s10096-004-1160-2. Epub 2004 Jun 30. PMID 15232720
- [Result] Mocroft A, Kirk O, Clumeck N, Gargalianos-Kakolyris P, Trocha H, Chentsova N, Antunes F, Stellbrink HJ, Phillips AN, Lundgren JD. The changing pattern of Kaposi sarcoma in patients with HIV, 1994-2003: the EuroSIDA Study. Cancer. 2004 Jun 15;100(12):2644-54. doi: 10.1002/cncr.20309. PMID 15197808
- [Result] Dragsted UB, Mocroft A, Vella S, Viard JP, Hansen AB, Panos G, Mercey D, Machala L, Horban A, Lundgren JD; EuroSIDA study group. Predictors of immunological failure after initial response to highly active antiretroviral therapy in HIV-1-infected adults: a EuroSIDA study. J Infect Dis. 2004 Jul 1;190(1):148-55. doi: 10.1086/420786. Epub 2004 Jun 9. PMID 15195254
- [Result] d'Arminio Monforte A, Cinque P, Mocroft A, Goebel FD, Antunes F, Katlama C, Justesen US, Vella S, Kirk O, Lundgren J; EuroSIDA Study Group. Changing incidence of central nervous system diseases in the EuroSIDA cohort. Ann Neurol. 2004 Mar;55(3):320-8. doi: 10.1002/ana.10827. PMID 14991809
- [Result] Blasko M. [EuroSIDA Study: downward trend of AIDS cases and AIDS mortality]. Dtsch Med Wochenschr. 2003 Sep 5;128(36):1814. No abstract available. German. PMID 14518432
- [Result] Florence E, Lundgren J, Dreezen C, Fisher M, Kirk O, Blaxhult A, Panos G, Katlama C, Vella S, Phillips A; EuroSIDA Study Group. Factors associated with a reduced CD4 lymphocyte count response to HAART despite full viral suppression in the EuroSIDA study. HIV Med. 2003 Jul;4(3):255-62. doi: 10.1046/j.1468-1293.2003.00156.x. PMID 12859325
- [Result] Mocroft A, Ledergerber B, Katlama C, Kirk O, Reiss P, d'Arminio Monforte A, Knysz B, Dietrich M, Phillips AN, Lundgren JD; EuroSIDA study group. Decline in the AIDS and death rates in the EuroSIDA study: an observational study. Lancet. 2003 Jul 5;362(9377):22-9. doi: 10.1016/s0140-6736(03)13802-0. PMID 12853195
- [Result] Mocroft A, Brettle R, Kirk O, Blaxhult A, Parkin JM, Antunes F, Francioli P, D'Arminio Monforte A, Fox Z, Lundgren JD; EuroSIDA study group. Changes in the cause of death among HIV positive subjects across Europe: results from the EuroSIDA study. AIDS. 2002 Aug 16;16(12):1663-71. doi: 10.1097/00002030-200208160-00012. PMID 12172088
- [Result] Mocroft A, Phillips AN, Friis-Moller N, Colebunders R, Johnson AM, Hirschel B, Saint-Marc T, Staub T, Clotet B, Lundgren JD; EuroSIDA study group. Response to antiretroviral therapy among patients exposed to three classes of antiretrovirals: results from the EuroSIDA study. Antivir Ther. 2002 Mar;7(1):21-30. PMID 12008784
- [Result] Lundgren JD, Mocroft A, Gatell JM, Ledergerber B, D'Arminio Monforte A, Hermans P, Goebel FD, Blaxhult A, Kirk O, Phillips AN; EuroSIDA Study Group. A clinically prognostic scoring system for patients receiving highly active antiretroviral therapy: results from the EuroSIDA study. J Infect Dis. 2002 Jan 15;185(2):178-87. doi: 10.1086/338267. Epub 2002 Jan 3. PMID 11807691
- [Result] Blaxhult A, Mocroft A, Phillips A, van Lunzen J, Bentwich Z, Stergiou G, Colebunders R, Benfield TL, Mulcahy F, Lundgren JD. Does European or non-European origin influence health care and prognosis for HIV patients in Europe? The EuroSIDA Study Group. HIV Med. 1999 Oct;1(1):2-9. doi: 10.1046/j.1468-1293.1999.00002.x. PMID 11737323
- [Result] Viard JP, Mocroft A, Chiesi A, Kirk O, Roge B, Panos G, Vetter N, Bruun JN, Johnson M, Lundgren JD; EuroSIDA Study Group. Influence of age on CD4 cell recovery in human immunodeficiency virus-infected patients receiving highly active antiretroviral therapy: evidence from the EuroSIDA study. J Infect Dis. 2001 Apr 15;183(8):1290-4. doi: 10.1086/319678. Epub 2001 Mar 26. PMID 11262215
- [Result] Mocroft A, Phillips AN, Miller V, Gatell J, van Lunzen J, Parkin JM, Weber R, Roge B, Lazzarin A, Lundgren JD; EuroSIDA study group. The use of and response to second-line protease inhibitor regimens: results from the EuroSIDA study. AIDS. 2001 Jan 26;15(2):201-9. doi: 10.1097/00002030-200101260-00009. PMID 11216928
- [Result] Mocroft A, Katlama C, Johnson AM, Pradier C, Antunes F, Mulcahy F, Chiesi A, Phillips AN, Kirk O, Lundgren JD. AIDS across Europe, 1994-98: the EuroSIDA study. Lancet. 2000 Jul 22;356(9226):291-6. doi: 10.1016/s0140-6736(00)02504-6. PMID 11071184
- [Result] Kirk O, Gatell JM, Mocroft A, Pedersen C, Proenca R, Brettle RP, Barton SE, Sudre P, Phillips AN. Infections with Mycobacterium tuberculosis and Mycobacterium avium among HIV-infected patients after the introduction of highly active antiretroviral therapy. EuroSIDA Study Group JD. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):865-72. doi: 10.1164/ajrccm.162.3.9908018. PMID 10988097
- [Result] Mocroft A, Miller V, Chiesi A, Blaxhult A, Katlama C, Clotet B, Barton S, Lundgren JD. Virological failure among patients on HAART from across Europe: results from the EuroSIDA study. Antivir Ther. 2000 Jun;5(2):107-12. PMID 10971863
- [Result] Paredes R, Mocroft A, Kirk O, Lazzarin A, Barton SE, van Lunzen J, Katzenstein TL, Antunes F, Lundgren JD, Clotet B. Predictors of virological success and ensuing failure in HIV-positive patients starting highly active antiretroviral therapy in Europe: results from the EuroSIDA study. Arch Intern Med. 2000 Apr 24;160(8):1123-32. doi: 10.1001/archinte.160.8.1123. PMID 10789605
- [Result] Mocroft A, Madge S, Johnson AM, Lazzarin A, Clumeck N, Goebel FD, Viard JP, Gatell J, Blaxhult A, Lundgren JD. A comparison of exposure groups in the EuroSIDA study: starting highly active antiretroviral therapy (HAART), response to HAART, and survival. J Acquir Immune Defic Syndr. 1999 Dec 1;22(4):369-78. doi: 10.1097/00126334-199912010-00008. PMID 10634199
- [Result] Chiesi A, Mocroft A, Dally LG, Miller V, Katlama C, Ledergerber B, Pedersen C, Phillips AN, Arcieri R, Lundgren JD. Regional survival differences across Europe in HIV-positive people: the EuroSIDA study. AIDS. 1999 Nov 12;13(16):2281-8. doi: 10.1097/00002030-199911120-00010. PMID 10563713
- [Result] Phillips AN, Grabar S, Tassie JM, Costagliola D, Lundgren JD, Egger M. Use of observational databases to evaluate the effectiveness of antiretroviral therapy for HIV infection: comparison of cohort studies with randomized trials. EuroSIDA, the French Hospital Database on HIV and the Swiss HIV Cohort Study Groups. AIDS. 1999 Oct 22;13(15):2075-82. doi: 10.1097/00002030-199910220-00010. PMID 10546860
- [Result] Mocroft A, Kirk O, Barton SE, Dietrich M, Proenca R, Colebunders R, Pradier C, dArminio Monforte A, Ledergerber B, Lundgren JD. Anaemia is an independent predictive marker for clinical prognosis in HIV-infected patients from across Europe. EuroSIDA study group. AIDS. 1999 May 28;13(8):943-50. doi: 10.1097/00002030-199905280-00010. PMID 10371175
- [Result] Weverling GJ, Mocroft A, Ledergerber B, Kirk O, Gonzales-Lahoz J, d'Arminio Monforte A, Proenca R, Phillips AN, Lundgren JD, Reiss P. Discontinuation of Pneumocystis carinii pneumonia prophylaxis after start of highly active antiretroviral therapy in HIV-1 infection. EuroSIDA Study Group. Lancet. 1999 Apr 17;353(9161):1293-8. doi: 10.1016/s0140-6736(99)03287-0. PMID 10218526
- [Result] Miller V, Mocroft A, Reiss P, Katlama C, Papadopoulos AI, Katzenstein T, van Lunzen J, Antunes F, Phillips AN, Lundgren JD. Relations among CD4 lymphocyte count nadir, antiretroviral therapy, and HIV-1 disease progression: results from the EuroSIDA study. Ann Intern Med. 1999 Apr 6;130(7):570-7. doi: 10.7326/0003-4819-130-7-199904060-00005. PMID 10189326
- [Result] Mocroft A, Vella S, Benfield TL, Chiesi A, Miller V, Gargalianos P, d'Arminio Monforte A, Yust I, Bruun JN, Phillips AN, Lundgren JD. Changing patterns of mortality across Europe in patients infected with HIV-1. EuroSIDA Study Group. Lancet. 1998 Nov 28;352(9142):1725-30. doi: 10.1016/s0140-6736(98)03201-2. PMID 9848347
- [Result] Kirk O, Mocroft A, Katzenstein TL, Lazzarin A, Antunes F, Francioli P, Brettle RP, Parkin JM, Gonzales-Lahoz J, Lundgren JD. Changes in use of antiretroviral therapy in regions of Europe over time. EuroSIDA Study Group. AIDS. 1998 Oct 22;12(15):2031-9. doi: 10.1097/00002030-199815000-00015. PMID 9814872
- [Result] Phillips AN, Katlama C, Barton S, Vella S, Blaxhult A, Clotet B, Goebel FD, Hirschel B, Pedersen C, Lundgren JD. Survival in 2367 zidovudine-treated patients according to use of other nucleoside analogue drugs. The EuroSIDA Study Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Mar 1;17(3):239-44. doi: 10.1097/00042560-199803010-00009. PMID 9495224
- [Result] Lundgren JD, Phillips AN, Vella S, Katlama C, Ledergerber B, Johnson AM, Reiss P, Gatell J, Clumeck N, Dietrich M, Benfield TL, Nielsen JO, Pedersen C. Regional differences in use of antiretroviral agents and primary prophylaxis in 3122 European HIV-infected patients. EuroSIDA Study Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Nov 1;16(3):153-60. doi: 10.1097/00042560-199711010-00003. PMID 9390566
- [Result] Vingerhoets J, Calvez V, Flandre P, Marcelin AG, Ceccherini-Silberstein F, Perno CF, Mercedes Santoro M, Bateson R, Nelson M, Cozzi-Lepri A, Grarup J, Lundgren J, Incardona F, Kaiser R, Sonnerborg A, Clotet B, Paredes R, Gunthard HF, Ledergerber B, Hoogstoel A, Nijs S, Tambuyzer L, Lavreys L, Opsomer M; Etravirine Cohort Study Group. Efficacy of etravirine combined with darunavir or other ritonavir-boosted protease inhibitors in HIV-1-infected patients: an observational study using pooled European cohort data. HIV Med. 2015 May;16(5):297-306. doi: 10.1111/hiv.12218. Epub 2015 Jan 14. PMID 25585664
- [Result] Marzolini C, Sabin C, Raffi F, Siccardi M, Mussini C, Launay O, Burger D, Roca B, Fehr J, Bonora S, Mocroft A, Obel N, Dauchy FA, Zangerle R, Gogos C, Gianotti N, Ammassari A, Torti C, Ghosn J, Chene G, Grarup J, Battegay M; Efavirenz, Obesity Project Team on behalf of Collaboration of Observational HIV Epidemiological Research Europe (COHERE) in EuroCoord. Impact of body weight on virological and immunological responses to efavirenz-containing regimens in HIV-infected, treatment-naive adults. AIDS. 2015 Jan 14;29(2):193-200. doi: 10.1097/QAD.0000000000000530. PMID 25426810
- [Result] Antiretroviral Therapy Cohort Collaboration (ART-CC); Vandenhende MA, Ingle S, May M, Chene G, Zangerle R, Van Sighem A, Gill MJ, Schwarze-Zander C, Hernandez-Novoa B, Obel N, Kirk O, Abgrall S, Guest J, Samji H, D'Arminio Monforte A, Llibre JM, Smith C, Cavassini M, Burkholder GA, Shepherd B, Crane HM, Sterne J, Morlat P. Impact of low-level viremia on clinical and virological outcomes in treated HIV-1-infected patients. AIDS. 2015 Jan 28;29(3):373-83. doi: 10.1097/QAD.0000000000000544. PMID 25686685
- [Result] Boesecke C, Grint D, Soriano V, Lundgren JD, d'Arminio Monforte A, Mitsura VM, Chentsova N, Hadziosmanovic V, Kirk O, Mocroft A, Peters L, Rockstroh JK; EuroSIDA in EuroCoord. Hepatitis C seroconversions in HIV infection across Europe: which regions and patient groups are affected? Liver Int. 2015 Nov;35(11):2384-91. doi: 10.1111/liv.12848. Epub 2015 Apr 29. PMID 25875966
- [Result] Bruyand M, Ryom L, Shepherd L, Fatkenheuer G, Grulich A, Reiss P, de Wit S, D Arminio Monforte A, Furrer H, Pradier C, Lundgren J, Sabin C; D:A:D study group. Cancer risk and use of protease inhibitor or nonnucleoside reverse transcriptase inhibitor-based combination antiretroviral therapy: the D: A: D study. J Acquir Immune Defic Syndr. 2015 Apr 15;68(5):568-77. doi: 10.1097/QAI.0000000000000523. PMID 25763785
- [Result] Mocroft A, Lundgren JD, Ross M, Law M, Reiss P, Kirk O, Smith C, Wentworth D, Neuhaus J, Fux CA, Moranne O, Morlat P, Johnson MA, Ryom L; D:A:D study group; Royal Free Hospital Clinic Cohort; INSIGHT study group; SMART study group; ESPRIT study group. Development and validation of a risk score for chronic kidney disease in HIV infection using prospective cohort data from the D:A:D study. PLoS Med. 2015 Mar 31;12(3):e1001809. doi: 10.1371/journal.pmed.1001809. eCollection 2015 Mar. PMID 25826420
- [Result] Friis-Moller N, Ryom L, Smith C, Weber R, Reiss P, Dabis F, De Wit S, Monforte AD, Kirk O, Fontas E, Sabin C, Phillips A, Lundgren J, Law M; D:A:D study group. An updated prediction model of the global risk of cardiovascular disease in HIV-positive persons: The Data-collection on Adverse Effects of Anti-HIV Drugs (D:A:D) study. Eur J Prev Cardiol. 2016 Jan;23(2):214-23. doi: 10.1177/2047487315579291. Epub 2015 Apr 16. PMID 25882821
- [Result] Mansfeld M, Skrahina A, Shepherd L, Schultze A, Panteleev AM, Miller RF, Miro JM, Zeltina I, Tetradov S, Furrer H, Kirk O, Grzeszczuk A, Bolokadze N, Matteelli A, Post FA, Lundgren JD, Mocroft A, Efsen A, Podlekareva DN; TB:HIV study group in EuroCoord. Major differences in organization and availability of health care and medicines for HIV/TB coinfected patients across Europe. HIV Med. 2015 Oct;16(9):544-52. doi: 10.1111/hiv.12256. Epub 2015 May 11. PMID 25959854
- [Result] Schultze A, Phillips AN, Paredes R, Battegay M, Rockstroh JK, Machala L, Tomazic J, Girard PM, Januskevica I, Gronborg-Laut K, Lundgren JD, Cozzi-Lepri A; EuroSIDA in EuroCOORD. HIV resistance testing and detected drug resistance in Europe. AIDS. 2015 Jul 17;29(11):1379-89. doi: 10.1097/QAD.0000000000000708. PMID 26091300
- [Result] Achhra AC, Mocroft A, Reiss P, Sabin C, Ryom L, de Wit S, Smith CJ, d'Arminio Monforte A, Phillips A, Weber R, Lundgren J, Law MG; D:A:D Study Group. Short-term weight gain after antiretroviral therapy initiation and subsequent risk of cardiovascular disease and diabetes: the D:A:D study. HIV Med. 2016 Apr;17(4):255-68. doi: 10.1111/hiv.12294. Epub 2015 Jul 28. PMID 26216031
- [Result] Grint D, Peters L, Rockstroh JK, Rakmanova A, Trofimova T, Lacombe K, Karpov I, Galli M, Domingo P, Kirk O, Lundgren JD, Mocroft A; EuroSIDA in EuroCoord. Liver-related death among HIV/hepatitis C virus-co-infected individuals: implications for the era of directly acting antivirals. AIDS. 2015 Jun 19;29(10):1205-15. doi: 10.1097/QAD.0000000000000674. PMID 25870984
- [Result] Podlekareva DN, Panteleev AM, Grint D, Post FA, Miro JM, Bruyand M, Furrer H, Obel N, Girardi E, Vasilenko A, Losso MH, Arenas-Pinto A, Cayla J, Rakhmanova A, Zeltina I, Werlinrud AM, Lundgren JD, Mocroft A, Kirk O; HIV/TB study group. Short- and long-term mortality and causes of death in HIV/tuberculosis patients in Europe. Eur Respir J. 2014 Jan;43(1):166-77. doi: 10.1183/09031936.00138712. Epub 2013 Jun 13. PMID 23766333
- [Result] Ryom L, Mocroft A, Kirk O, Ross M, Reiss P, Fux CA, Morlat P, Moranne O, Smith C, El-Sadr W, Law M, Lundgren JD. Predictors of advanced chronic kidney disease and end-stage renal disease in HIV-positive persons. AIDS. 2014 Jan 14;28(2):187-99. doi: 10.1097/QAD.0000000000000042. PMID 24361680
- [Result] Zoufaly A, Cozzi-Lepri A, Reekie J, Kirk O, Lundgren J, Reiss P, Jevtovic D, Machala L, Zangerle R, Mocroft A, Van Lunzen J; EuroSIDA in EuroCoord. Immuno-virological discordance and the risk of non-AIDS and AIDS events in a large observational cohort of HIV-patients in Europe. PLoS One. 2014 Jan 31;9(1):e87160. doi: 10.1371/journal.pone.0087160. eCollection 2014. PMID 24498036
- [Result] Grint D, Peters L, Rockstroh JK, de Wit S, Mitsura VM, Knysz B, Pedersen C, Kirk O, Lundgren JD, Mocroft A; EuroSIDA in EuroCoord. Increased incidence of antiretroviral drug discontinuation among patients with viremic hepatitis C virus coinfection and high hyaluronic acid, a marker of liver fibrosis. AIDS. 2014 Feb 20;28(4):577-87. doi: 10.1097/QAD.0000000000000069. PMID 24468998
- [Result] Mocroft A, Ryom L, Reiss P, Furrer H, D'Arminio Monforte A, Gatell J, de Wit S, Beniowski M, Lundgren JD, Kirk O; EuroSIDA in EuroCOORD. A comparison of estimated glomerular filtration rates using Cockcroft-Gault and the Chronic Kidney Disease Epidemiology Collaboration estimating equations in HIV infection. HIV Med. 2014 Mar;15(3):144-52. doi: 10.1111/hiv.12095. Epub 2013 Oct 3. PMID 24118916
- [Result] Shepherd L, Souberbielle JC, Bastard JP, Fellahi S, Capeau J, Reekie J, Reiss P, Blaxhult A, Bickel M, Leen C, Kirk O, Lundgren JD, Mocroft A, Viard JP; EuroSIDA in EuroCOORD. Prognostic value of vitamin D level for all-cause mortality, and association with inflammatory markers, in HIV-infected persons. J Infect Dis. 2014 Jul 15;210(2):234-43. doi: 10.1093/infdis/jiu074. Epub 2014 Feb 3. PMID 24493824
- [Result] Mocroft A, Ryom L, Begovac J, Monforte AD, Vassilenko A, Gatell J, Florence E, Ormaasen V, Kirk O, Lundgren JD; EuroSIDA in EuroCOORD. Deteriorating renal function and clinical outcomes in HIV-positive persons. AIDS. 2014 Mar 13;28(5):727-37. doi: 10.1097/QAD.0000000000000134. PMID 24983543
- [Result] Kamara DA, Ryom L, Ross M, Kirk O, Reiss P, Morlat P, Moranne O, Fux CA, Mocroft A, Sabin C, Lundgren JD, Smith CJ; D:A:D study Group. Development of a definition for Rapid Progression (RP) of renal function in HIV-positive persons: the D:A:D study. BMC Nephrol. 2014 Mar 25;15:51. doi: 10.1186/1471-2369-15-51. PMID 24666792
- [Result] Engsig FN, Zangerle R, Katsarou O, Dabis F, Reiss P, Gill J, Porter K, Sabin C, Riordan A, Fatkenheuer G, Gutierrez F, Raffi F, Kirk O, Mary-Krause M, Stephan C, de Olalla PG, Guest J, Samji H, Castagna A, d'Arminio Monforte A, Skaletz-Rorowski A, Ramos J, Lapadula G, Mussini C, Force L, Meyer L, Lampe F, Boufassa F, Bucher HC, De Wit S, Burkholder GA, Teira R, Justice AC, Sterling TR, M Crane H, Gerstoft J, Grarup J, May M, Chene G, Ingle SM, Sterne J, Obel N; Antiretroviral Therapy Cohort Collaboration (ART-CC) and the Collaboration of Observational HIV Epidemiological Research Europe (COHERE) in EuroCoord. Long-term mortality in HIV-positive individuals virally suppressed for >3 years with incomplete CD4 recovery. Clin Infect Dis. 2014 May;58(9):1312-21. doi: 10.1093/cid/ciu038. Epub 2014 Jan 22. PMID 24457342
- [Result] Petoumenos K, Reiss P, Ryom L, Rickenbach M, Sabin CA, El-Sadr W, d'Arminio Monforte A, Phillips AN, De Wit S, Kirk O, Dabis F, Pradier C, Lundgren JD, Law MG; D:A:D study group. Increased risk of cardiovascular disease (CVD) with age in HIV-positive men: a comparison of the D:A:D CVD risk equation and general population CVD risk equations. HIV Med. 2014 Nov;15(10):595-603. doi: 10.1111/hiv.12162. Epub 2014 May 19. PMID 24840675
- [Result] Peters L, Mocroft A, Soriano V, Rockstroh JK, Kirkby N, Reiss P, Katlama C, Zakharova N, Flisiak R, Lundgren JD; EuroSIDA in EuroCoord. High rate of hepatitis C virus (HCV) recurrence in HIV-infected individuals with spontaneous HCV RNA clearance. HIV Med. 2014 Nov;15(10):615-20. doi: 10.1111/hiv.12160. Epub 2014 May 11. PMID 24814468
- [Result] Natural History Project Working Group for the Collaboration of Observational HIV Epidemiological Research Europe (COHERE) in EuroCoord. Factors associated with short-term changes in HIV viral load and CD4(+) cell count in antiretroviral-naive individuals. AIDS. 2014 Jun 1;28(9):1351-6. doi: 10.1097/QAD.0000000000000224. PMID 24959963
- [Result] Ingle SM, May MT, Gill MJ, Mugavero MJ, Lewden C, Abgrall S, Fatkenheuer G, Reiss P, Saag MS, Manzardo C, Grabar S, Bruyand M, Moore D, Mocroft A, Sterling TR, D'Arminio Monforte A, Hernando V, Teira R, Guest J, Cavassini M, Crane HM, Sterne JA; Antiretroviral Therapy Cohort Collaboration. Impact of risk factors for specific causes of death in the first and subsequent years of antiretroviral therapy among HIV-infected patients. Clin Infect Dis. 2014 Jul 15;59(2):287-97. doi: 10.1093/cid/ciu261. Epub 2014 Apr 24. PMID 24771333
- [Result] Smith CJ, Ryom L, Weber R, Morlat P, Pradier C, Reiss P, Kowalska JD, de Wit S, Law M, el Sadr W, Kirk O, Friis-Moller N, Monforte Ad, Phillips AN, Sabin CA, Lundgren JD; D:A:D Study Group. Trends in underlying causes of death in people with HIV from 1999 to 2011 (D:A:D): a multicohort collaboration. Lancet. 2014 Jul 19;384(9939):241-8. doi: 10.1016/S0140-6736(14)60604-8. PMID 25042234
- [Result] Mocroft A, Reiss P, Rakhmanova A, Banhegyi D, Phillips AN, De Wit S, Ristola M, Lundgren JD, Grarup J, Kirk O; EuroSIDA in EuroCOORD. A survey of ATRIPLA use in clinical practice as first-line therapy in HIV-positive persons in Europe. Infection. 2014 Aug;42(4):757-62. doi: 10.1007/s15010-014-0630-4. Epub 2014 Jun 6. PMID 24902520
- [Result] Socio-economic Inequalities and HIV Writing Group for Collaboration of Observational HIV Epidemiological Research in Europe (COHERE) in EuroCoord; Lodi S, Dray-Spira R, Touloumi G, Braun D, Teira R, D'Arminio Monforte A, Gallois A, Zangerle R, Spire B, Dabis F, Stahelin C, Termote M, Kirk O, Chene G, Egger M, del Amo J. Delayed HIV diagnosis and initiation of antiretroviral therapy: inequalities by educational level, COHERE in EuroCoord. AIDS. 2014 Sep 24;28(15):2297-306. doi: 10.1097/QAD.0000000000000410. PMID 25313585
- [Result] Klein MB, Young J, Dunn D, Ledergerber B, Sabin C, Cozzi-Lepri A, Dabis F, Harrigan R, Tan DH, Walmsley S, Gill J, Cooper C, Scherrer AU, Mocroft A, Hogg RS, Smaill F; Canadian-European Clade Collaboration. The effects of HIV-1 subtype and ethnicity on the rate of CD4 cell count decline in patients naive to antiretroviral therapy: a Canadian-European collaborative retrospective cohort study. CMAJ Open. 2014 Oct 1;2(4):E318-29. doi: 10.9778/cmajo.20140017. eCollection 2014 Oct. PMID 25485259
- [Result] Borges AH, Lundgren JD, Ridolfo A, Katlama C, Antunes F, Grzeszczuk A, Blaxhult A, Mitsura VM, Doroana M, Battegay M, Gargalianos P, Mocroft A; EuroSIDA in EuroCOORD. Thrombocytopenia is associated with an increased risk of cancer during treated HIV disease. AIDS. 2014 Nov 13;28(17):2565-71. doi: 10.1097/QAD.0000000000000433. PMID 25574959
- [Result] Cozzi-Lepri A, Noguera-Julian M, Di Giallonardo F, Schuurman R, Daumer M, Aitken S, Ceccherini-Silberstein F, D'Arminio Monforte A, Geretti AM, Booth CL, Kaiser R, Michalik C, Jansen K, Masquelier B, Bellecave P, Kouyos RD, Castro E, Furrer H, Schultze A, Gunthard HF, Brun-Vezinet F, Paredes R, Metzner KJ; CHAIN Minority HIV-1 Variants Working Group. Low-frequency drug-resistant HIV-1 and risk of virological failure to first-line NNRTI-based ART: a multicohort European case-control study using centralized ultrasensitive 454 pyrosequencing. J Antimicrob Chemother. 2015 Mar;70(3):930-40. doi: 10.1093/jac/dku426. Epub 2014 Oct 21. PMID 25336166
- [Result] Sogaard OS, Reekie J, Ristola M, Jevtovic D, Karpov I, Beniowski M, Servitskiy S, Domingo P, Reiss P, Mocroft A, Kirk O. Severe bacterial non-aids infections in HIV-positive persons: incidence rates and risk factors. J Infect. 2013 May;66(5):439-46. doi: 10.1016/j.jinf.2012.12.012. Epub 2013 Jan 24. PMID 23353671
- [Result] Monforte Ad, Reiss P, Ryom L, El-Sadr W, Dabis F, De Wit S, Worm SW, Law MG, Weber R, Kirk O, Pradier C, Phillips AN, Lundgren JD, Sabin CA. Atazanavir is not associated with an increased risk of cardio- or cerebrovascular disease events. AIDS. 2013 Jan 28;27(3):407-15. doi: 10.1097/QAD.0b013e32835b2ef1. PMID 23291539
- [Result] Tate JP, Justice AC, Hughes MD, Bonnet F, Reiss P, Mocroft A, Nattermann J, Lampe FC, Bucher HC, Sterling TR, Crane HM, Kitahata MM, May M, Sterne JA. An internationally generalizable risk index for mortality after one year of antiretroviral therapy. AIDS. 2013 Feb 20;27(4):563-72. doi: 10.1097/QAD.0b013e32835b8c7f. PMID 23095314
- [Result] Podlekareva DN, Grint D, Post FA, Mocroft A, Panteleev AM, Miller RF, Miro JM, Bruyand M, Furrer H, Riekstina V, Girardi E, Losso MH, Cayla JA, Malashenkov EA, Obel N, Skrahina AM, Lundgren JD, Kirk O; HIV-TB Study Group. Health care index score and risk of death following tuberculosis diagnosis in HIV-positive patients. Int J Tuberc Lung Dis. 2013 Feb;17(2):198-206. doi: 10.5588/ijtld.12.0224. PMID 23317955
- [Result] Pursuing Later Treatment Option II (PLATO II) Project Team of the Collaboration of Observational HIV Epidemiological Research Europe (COHERE); Costagliola D, Ledergerber B, Torti C, van Sighem A, Podzamczer D, Mocroft A, Dorrucci M, Masquelier B, de Luca A, Jansen K, De Wit S, Obel N, Fatkenheuer G, Touloumi G, Mussini C, Castagna A, Stephan C, Garcia F, Zangerle R, Duval X, Perez-Hoyos S, Meyer L, Ghosn J, Fabre-Colin C, Kjaer J, Chene G, Grarup J, Phillips A, Lodwick R, Torti C, Dorrucci M, Gunthard HF, Michalik C, Chrysos G, Castagna A. Predictors of CD4(+) T-cell counts of HIV type 1-infected persons after virologic failure of all 3 original antiretroviral drug classes. J Infect Dis. 2013 Mar 1;207(5):759-67. doi: 10.1093/infdis/jis752. Epub 2012 Dec 7. PMID 23225900
- [Result] Abgrall S, Ingle SM, May MT, Costagliola D, Mercie P, Cavassini M, Reekie J, Samji H, Gill MJ, Crane HM, Tate J, Sterling TR, Antinori A, Reiss P, Saag MS, Mugavero MJ, Phillips A, Manzardo C, Wasmuth JC, Stephan C, Guest JL, Gomez Sirvent JL, Sterne JA; Antiretroviral Therapy Cohort Collaboration (ART-CC). Durability of first ART regimen and risk factors for modification, interruption or death in HIV-positive patients starting ART in Europe and North America 2002-2009. AIDS. 2013 Mar 13;27(5):803-13. doi: 10.1097/QAD.0b013e32835cb997. PMID 23719350
- [Result] Sabin CA, Ryom L, Kovari H, Kirk O, de Wit S, Law M, Reiss P, Dabis F, Pradier C, El-Sadr W, Monforte Ad, Kamara D, Phillips AN, Lundgren JD. Association between ALT level and the rate of cardio/cerebrovascular events in HIV-positive individuals: the D: A: D study. J Acquir Immune Defic Syndr. 2013 Aug 1;63(4):456-63. doi: 10.1097/QAI.0b013e318291cd29. PMID 23535291
- [Result] Grint D, Peters L, Reekie J, Soriano V, Kirk O, Knysz B, Suetnov O, Lazzarin A, Ledergerber B, Rockstroh JK, Mocroft A; EuroSIDA in EuroCoord (European Coordinating Committee for the Integration of Ongoing Coordination Actions Related to Clinical and Epidemiological HIV Research). Stability of hepatitis C virus (HCV) RNA levels among interferon-naive HIV/HCV-coinfected individuals treated with combination antiretroviral therapy. HIV Med. 2013 Jul;14(6):370-8. doi: 10.1111/hiv.12033. Epub 2013 Mar 27. PMID 23534815
- [Result] Mocroft A, Phillips AN, Gatell J, Horban A, Ledergerber B, Zilmer K, Jevtovic D, Maltez F, Podlekareva D, Lundgren JD; EuroSIDA study in EuroCOORD. CD4 cell count and viral load-specific rates of AIDS, non-AIDS and deaths according to current antiretroviral use. AIDS. 2013 Mar 27;27(6):907-918. doi: 10.1097/QAD.0b013e32835cb766. PMID 23698060
- [Result] Rockstroh JK, Peters L, Grint D, Soriano V, Reiss P, Monforte Ad, Beniowski M, Losso MH, Kirk O, Kupfer B, Mocroft A; EuroSIDA in EuroCoord. Does hepatitis C viremia or genotype predict the risk of mortality in individuals co-infected with HIV? J Hepatol. 2013 Aug;59(2):213-20. doi: 10.1016/j.jhep.2013.04.005. Epub 2013 Apr 11. PMID 23583272
- [Result] Ryom L, Kirk O, Lundgren JD, Reiss P, Pedersen C, De Wit S, Buzunova S, Gasiorowski J, Gatell JM, Mocroft A; EuroSIDA in EuroCoord. Advanced chronic kidney disease, end-stage renal disease and renal death among HIV-positive individuals in Europe. HIV Med. 2013 Sep;14(8):503-8. doi: 10.1111/hiv.12038. Epub 2013 Apr 16. PMID 23590641
- [Result] Ryom L, Mocroft A, Kirk O, Worm SW, Kamara DA, Reiss P, Ross M, Fux CA, Morlat P, Moranne O, Smith C, Lundgren JD; D:A:D Study Group. Association between antiretroviral exposure and renal impairment among HIV-positive persons with normal baseline renal function: the D:A:D study. J Infect Dis. 2013 May 1;207(9):1359-69. doi: 10.1093/infdis/jit043. Epub 2013 Feb 4. PMID 23382571
- [Result] Peters L, Mocroft A, Soriano V, Rockstroh J, Rauch A, Karlsson A, Knysz B, Pradier C, Zilmer K, Lundgren JD; for EuroSIDA in EuroCoord. Hyaluronic acid levels predict risk of hepatic encephalopathy and liver-related death in HIV/viral hepatitis coinfected patients. PLoS One. 2013 May 27;8(5):e64283. doi: 10.1371/journal.pone.0064283. Print 2013. PMID 23724041
- [Result] Kovari H, Sabin CA, Ledergerber B, Ryom L, Worm SW, Smith C, Phillips A, Reiss P, Fontas E, Petoumenos K, De Wit S, Morlat P, Lundgren JD, Weber R. Antiretroviral drug-related liver mortality among HIV-positive persons in the absence of hepatitis B or C virus coinfection: the data collection on adverse events of anti-HIV drugs study. Clin Infect Dis. 2013 Mar;56(6):870-9. doi: 10.1093/cid/cis919. Epub 2012 Oct 22. PMID 23090925
- [Result] Mocroft A, Lundgren JD, Sabin ML, Monforte Ad, Brockmeyer N, Casabona J, Castagna A, Costagliola D, Dabis F, De Wit S, Fatkenheuer G, Furrer H, Johnson AM, Lazanas MK, Leport C, Moreno S, Obel N, Post FA, Reekie J, Reiss P, Sabin C, Skaletz-Rorowski A, Suarez-Lozano I, Torti C, Warszawski J, Zangerle R, Fabre-Colin C, Kjaer J, Chene G, Grarup J, Kirk O; Collaboration of Observational HIV Epidemiological Research Europe (COHERE) study in EuroCoord. Risk factors and outcomes for late presentation for HIV-positive persons in Europe: results from the Collaboration of Observational HIV Epidemiological Research Europe Study (COHERE). PLoS Med. 2013;10(9):e1001510. doi: 10.1371/journal.pmed.1001510. Epub 2013 Sep 3. PMID 24137103
- [Result] Kaulich-Bartz J, Dam W, May MT, Lederberger B, Widmer U, Phillips AN, Grabar S, Mocroft A, Vilaro J, van Sighem A, Moreno S, Dabis F, Monforte AD, Teira R, Ingle SM, Sterne JA; Writing Committee for the Antiretroviral Therapy Cohort Collaboration. Insurability of HIV-positive people treated with antiretroviral therapy in Europe: collaborative analysis of HIV cohort studies. AIDS. 2013 Jun 19;27(10):1641-55. doi: 10.1097/QAD.0b013e3283601199. PMID 23449349
- [Result] Mocroft A, Furrer HJ, Miro JM, Reiss P, Mussini C, Kirk O, Abgrall S, Ayayi S, Bartmeyer B, Braun D, Castagna A, d'Arminio Monforte A, Gazzard B, Gutierrez F, Hurtado I, Jansen K, Meyer L, Munoz P, Obel N, Soler-Palacin P, Papadopoulos A, Raffi F, Ramos JT, Rockstroh JK, Salmon D, Torti C, Warszawski J, de Wit S, Zangerle R, Fabre-Colin C, Kjaer J, Chene G, Grarup J, Lundgren JD; Opportunistic Infections Working Group on behalf of the Collaboration of Observational HIV Epidemiological Research Europe (COHERE) study in EuroCOORD. The incidence of AIDS-defining illnesses at a current CD4 count >/= 200 cells/muL in the post-combination antiretroviral therapy era. Clin Infect Dis. 2013 Oct;57(7):1038-47. doi: 10.1093/cid/cit423. Epub 2013 Aug 6. PMID 23921881
- [Result] Worm SW, Bower M, Reiss P, Bonnet F, Law M, Fatkenheuer G, d'Arminio Monforte A, Abrams DI, Grulich A, Fontas E, Kirk O, Furrer H, De Wit S, Phillips A, Lundgren JD, Sabin CA; D:A:D Study Group. Non-AIDS defining cancers in the D:A:D Study--time trends and predictors of survival: a cohort study. BMC Infect Dis. 2013 Oct 9;13:471. doi: 10.1186/1471-2334-13-471. PMID 24106926
- [Result] May MT, Ingle SM, Costagliola D, Justice AC, de Wolf F, Cavassini M, D'Arminio Monforte A, Casabona J, Hogg RS, Mocroft A, Lampe FC, Dabis F, Fatkenheuer G, Sterling TR, del Amo J, Gill MJ, Crane HM, Saag MS, Guest J, Brodt HR, Sterne JA; Antiretroviral Cohort Collaboration. Cohort profile: Antiretroviral Therapy Cohort Collaboration (ART-CC). Int J Epidemiol. 2014 Jun;43(3):691-702. doi: 10.1093/ije/dyt010. Epub 2013 Apr 18. PMID 23599235
- [Result] Post FA, Grint D, Werlinrud AM, Panteleev A, Riekstina V, Malashenkov EA, Skrahina A, Duiculescu D, Podlekareva D, Karpov I, Bondarenko V, Chentsova N, Lundgren J, Mocroft A, Kirk O, Miro JM; HIV-TB Study Group. Multi-drug-resistant tuberculosis in HIV positive patients in Eastern Europe. J Infect. 2014 Mar;68(3):259-63. doi: 10.1016/j.jinf.2013.09.034. Epub 2013 Nov 16. PMID 24247067
- [Result] Efsen AM, Panteleev AM, Grint D, Podlekareva DN, Vassilenko A, Rakhmanova A, Zeltina I, Losso MH, Miller RF, Girardi E, Cayla J, Post FA, Miro JM, Bruyand M, Furrer H, Obel N, Lundgren JD, Mocroft A, Kirk O; HIV/TB Study Group. TB meningitis in HIV-positive patients in Europe and Argentina: clinical outcome and factors associated with mortality. Biomed Res Int. 2013;2013:373601. doi: 10.1155/2013/373601. Epub 2013 Dec 31. PMID 24699884
- [Result] Sabin CA, Ryom L, De Wit S, Mocroft A, Phillips AN, Worm SW, Weber R, D'Arminio Monforte A, Reiss P, Kamara D, El-Sadr W, Pradier C, Dabis F, Law M, Lundgren J; D:A:D Study Group. Associations between immune depression and cardiovascular events in HIV infection. AIDS. 2013 Nov 13;27(17):2735-48. doi: 10.1097/01.aids.0000432457.91228.f3. PMID 23842128
- [Result] Kowalska JD, Reekie J, Mocroft A, Reiss P, Ledergerber B, Gatell J, d'Arminio Monforte A, Phillips A, Lundgren JD, Kirk O; EuroSIDA study group. Long-term exposure to combination antiretroviral therapy and risk of death from specific causes: no evidence for any previously unidentified increased risk due to antiretroviral therapy. AIDS. 2012 Jan 28;26(3):315-23. doi: 10.1097/QAD.0b013e32834e8805. PMID 22112597
- [Result] Pursuing Later Treatment Option II (PLATO II) project team; Observational HIV Epidemiological Research Europe (COHERE) Group; Costagliola D, Lodwick R, Ledergerber B, Torti C, van Sighem A, Podzamczer D, Mocroft A, Dorrucci M, Masquelier B, de Luca A, Jansen K, De Wit S, Obel N, Fatkenheuer G, Touoloumi G, Mussini C, Castagna A, Stephan C, Garcia F, Zangerle R, Duval X, Perez-Hoyos S, Meyer L, Ghosn J, Fabre-Colin C, Kjaer J, Chene G, Grarup J, Phillips A. Trends in virological and clinical outcomes in individuals with HIV-1 infection and virological failure of drugs from three antiretroviral drug classes: a cohort study. Lancet Infect Dis. 2012 Feb;12(2):119-27. doi: 10.1016/S1473-3099(11)70248-1. Epub 2011 Oct 9. PMID 21988895
- [Result] Peters L, Grint D, Lundgren JD, Rockstroh JK, Soriano V, Reiss P, Grzeszczuk A, Sambatakou H, Mocroft A, Kirk O; EuroSIDA in EuroCoord. Hepatitis C virus viremia increases the incidence of chronic kidney disease in HIV-infected patients. AIDS. 2012 Sep 24;26(15):1917-26. doi: 10.1097/QAD.0b013e3283574e71. PMID 22781222
- [Result] Collaboration of Observational HIV Epidemiological Research Europe (COHERE) in EuroCoord; Lewden C, Bouteloup V, De Wit S, Sabin C, Mocroft A, Wasmuth JC, van Sighem A, Kirk O, Obel N, Panos G, Ghosn J, Dabis F, Mary-Krause M, Leport C, Perez-Hoyos S, Sobrino-Vegas P, Stephan C, Castagna A, Antinori A, d'Arminio Monforte A, Torti C, Mussini C, Isern V, Calmy A, Teira R, Egger M, Grarup J, Chene G. All-cause mortality in treated HIV-infected adults with CD4 >/=500/mm3 compared with the general population: evidence from a large European observational cohort collaboration. Int J Epidemiol. 2012 Apr;41(2):433-45. doi: 10.1093/ije/dyr164. Epub 2011 Nov 28. PMID 22493325
- [Result] Worm SW, Kamara DA, Reiss P, Fontas E, De Wit S, El-Sadr W, D'Arminio Monforte A, Law M, Phillips A, Ryom L, Dabis F, Weber R, Sabin C, Lundgren JD; D:A:D Study Group. Evaluation of HIV protease inhibitor use and the risk of sudden death or nonhemorrhagic stroke. J Infect Dis. 2012 Feb 15;205(4):535-9. doi: 10.1093/infdis/jir788. Epub 2012 Jan 5. PMID 22223855
- [Result] Petoumenos K, Worm SW, Fontas E, Weber R, De Wit S, Bruyand M, Reiss P, El-Sadr W, Monforte AD, Friis-Moller N, Lundgren JD, Law MG; D:A:D Study Group. Predicting the short-term risk of diabetes in HIV-positive patients: the Data Collection on Adverse Events of Anti-HIV Drugs (D:A:D) study. J Int AIDS Soc. 2012 Oct 10;15(2):17426. doi: 10.7448/IAS.15.2.17426. PMID 23078769
- [Result] Opportunistic Infections Project Team of the Collaboration of Observational HIV Epidemiological Research in Europe (COHERE) in EuroCoord; Young J, Psichogiou M, Meyer L, Ayayi S, Grabar S, Raffi F, Reiss P, Gazzard B, Sharland M, Gutierrez F, Obel N, Kirk O, Miro JM, Furrer H, Castagna A, De Wit S, Munoz J, Kjaer J, Grarup J, Chene G, Bucher H. CD4 cell count and the risk of AIDS or death in HIV-Infected adults on combination antiretroviral therapy with a suppressed viral load: a longitudinal cohort study from COHERE. PLoS Med. 2012;9(3):e1001194. doi: 10.1371/journal.pmed.1001194. Epub 2012 Mar 20. PMID 22448150
- [Result] Mocroft A, Bannister WP, Kirk O, Kowalska JD, Reiss P, D'Arminio-Monforte A, Gatell J, Fisher M, Trocha H, Rakhmanova A, Lundgren JD; EuroSIDA Study in EuroCOORD. The clinical benefits of antiretroviral therapy in severely immunocompromised HIV-1-infected patients with and without complete viral suppression. Antivir Ther. 2012;17(7):1291-300. doi: 10.3851/IMP2407. Epub 2012 Sep 26. PMID 23013779
- [Result] HCV working group of the Collaboration of Observational HIV Epidemiological Research in Europe (COHERE) in EuroCoord. Effect of hepatitis C treatment on CD4+ T-cell counts and the risk of death in HIV-HCV-coinfected patients: the COHERE collaboration. Antivir Ther. 2012;17(8):1541-50. doi: 10.3851/IMP2263. Epub 2012 Jul 24. PMID 22869294
- [Result] May MT, Hogg RS, Justice AC, Shepherd BE, Costagliola D, Ledergerber B, Thiebaut R, Gill MJ, Kirk O, van Sighem A, Saag MS, Navarro G, Sobrino-Vegas P, Lampe F, Ingle S, Guest JL, Crane HM, D'Arminio Monforte A, Vehreschild JJ, Sterne JA; Antiretroviral Therapy Cohort Collaboration (ART-CC). Heterogeneity in outcomes of treated HIV-positive patients in Europe and North America: relation with patient and cohort characteristics. Int J Epidemiol. 2012 Dec;41(6):1807-20. doi: 10.1093/ije/dys164. Epub 2012 Nov 12. PMID 23148105
- [Result] Murray M, Hogg RS, Lima VD, May MT, Moore DM, Abgrall S, Bruyand M, D'Arminio Monforte A, Tural C, Gill MJ, Harris RJ, Reiss P, Justice A, Kirk O, Saag M, Smith CJ, Weber R, Rockstroh J, Khaykin P, Sterne JA; Antiretroviral Therapy Cohort Collaboration (ART-CC). The effect of injecting drug use history on disease progression and death among HIV-positive individuals initiating combination antiretroviral therapy: collaborative cohort analysis. HIV Med. 2012 Feb;13(2):89-97. doi: 10.1111/j.1468-1293.2011.00940.x. Epub 2011 Aug 7. PMID 21819529
- [Result] Bannister WP, Cozzi-Lepri A, Kjaer J, Clotet B, Lazzarin A, Viard JP, Kronborg G, Duiculescu D, Beniowski M, Machala L, Phillips A; EuroSIDA group. Estimating prevalence of accumulated HIV-1 drug resistance in a cohort of patients on antiretroviral therapy. J Antimicrob Chemother. 2011 Apr;66(4):901-11. doi: 10.1093/jac/dkr006. Epub 2011 Jan 31. PMID 21393179
- [Result] Petoumenos K, Worm S, Reiss P, de Wit S, d'Arminio Monforte A, Sabin C, Friis-Moller N, Weber R, Mercie P, Pradier C, El-Sadr W, Kirk O, Lundgren J, Law M; D:A:D Study Group. Rates of cardiovascular disease following smoking cessation in patients with HIV infection: results from the D:A:D study(*). HIV Med. 2011 Aug;12(7):412-21. doi: 10.1111/j.1468-1293.2010.00901.x. Epub 2011 Jan 20. PMID 21251183
- [Result] Kruk A, Bannister W, Podlekareva DN, Chentsova NP, Rakhmanova AG, Horban A, Domingo P, Mocroft A, Lundgren JD, Kirk O; EuroSIDA study group. Tuberculosis among HIV-positive patients across Europe: changes over time and risk factors. AIDS. 2011 Jul 31;25(12):1505-13. doi: 10.1097/QAD.0b013e328348fafd. PMID 21610489
- [Result] Bohlius J, Schmidlin K, Boue F, Fatkenheuer G, May M, Caro-Murillo AM, Mocroft A, Bonnet F, Clifford G, Paparizos V, Miro JM, Obel N, Prins M, Chene G, Egger M; Collaboration of Observational HIV Epidemiological Research Europe. HIV-1-related Hodgkin lymphoma in the era of combination antiretroviral therapy: incidence and evolution of CD4(+) T-cell lymphocytes. Blood. 2011 Jun 9;117(23):6100-8. doi: 10.1182/blood-2010-08-301531. Epub 2011 Mar 2. PMID 21368291
- [Result] Kowalska JD, Friis-Moller N, Kirk O, Bannister W, Mocroft A, Sabin C, Reiss P, Gill J, Lewden C, Phillips A, D'Arminio Monforte A, Law M, Sterne J, De Wit S, Lundgren JD; CoDe Working Group; D:A:D Study Group. The Coding Causes of Death in HIV (CoDe) Project: initial results and evaluation of methodology. Epidemiology. 2011 Jul;22(4):516-23. doi: 10.1097/EDE.0b013e31821b5332. PMID 21522013
- [Result] Soriano V, Grint D, d'Arminio Monforte A, Horban A, Leen C, Poveda E, Antunes F, de Wit S, Lundgren J, Rockstroh J, Peters L. Hepatitis delta in HIV-infected individuals in Europe. AIDS. 2011 Oct 23;25(16):1987-92. doi: 10.1097/QAD.0b013e32834babb3. PMID 21857493
- [Result] Reekie J, Gatell JM, Yust I, Bakowska E, Rakhmanova A, Losso M, Krasnov M, Francioli P, Kowalska JD, Mocroft A; EuroSIDA in EuroCoord. Fatal and nonfatal AIDS and non-AIDS events in HIV-1-positive individuals with high CD4 cell counts according to viral load strata. AIDS. 2011 Nov 28;25(18):2259-68. doi: 10.1097/QAD.0b013e32834cdb4b. PMID 21918422
- [Result] Paredes R, Puertas MC, Bannister W, Kisic M, Cozzi-Lepri A, Pou C, Bellido R, Betancor G, Bogner J, Gargalianos P, Banhegyi D, Clotet B, Lundgren J, Menendez-Arias L, Martinez-Picado J; EuroSIDA Study Group. A376S in the connection subdomain of HIV-1 reverse transcriptase confers increased risk of virological failure to nevirapine therapy. J Infect Dis. 2011 Sep 1;204(5):741-52. doi: 10.1093/infdis/jir385. PMID 21844300
- [Result] Cozzi-Lepri A, Prosperi MC, Kjaer J, Dunn D, Paredes R, Sabin CA, Lundgren JD, Phillips AN, Pillay D; EuroSIDA Study; United Kingdom CHIC/United Kingdom HDRD Study. Can linear regression modeling help clinicians in the interpretation of genotypic resistance data? An application to derive a lopinavir-score. PLoS One. 2011;6(11):e25665. doi: 10.1371/journal.pone.0025665. Epub 2011 Nov 16. PMID 22110581
- [Result] Cozzi-Lepri A, Paredes, Phillips AN, Clotet B, Kjaer J, Von Wyl V, Kronborg G, Castagna A, Bogner JR, Lundgren JD; EuroSIDA in EuroCoord. The rate of accumulation of nonnucleoside reverse transcriptase inhibitor (NNRTI) resistance in patients kept on a virologically failing regimen containing an NNRTI*. HIV Med. 2012 Jan;13(1):62-72. doi: 10.1111/j.1468-1293.2011.00943.x. Epub 2011 Aug 17. PMID 21848790
- [Result] Worm SW, Kamara DA, Reiss P, Kirk O, El-Sadr W, Fux C, Fontas E, Phillips A, D'Arminio Monforte A, De Wit S, Petoumenos K, Friis-Mller N, Mercie P, Lundgren JD, Sabin C. Elevated triglycerides and risk of myocardial infarction in HIV-positive persons. AIDS. 2011 Jul 31;25(12):1497-504. doi: 10.1097/QAD.0b013e32834917c6. PMID 21633288
- [Result] Data Collection on Adverse Events of Anti-HIV Drugs (D:A:D) Study. The impact of fasting on the interpretation of triglyceride levels for predicting myocardial infarction risk in HIV-positive individuals: the D:A:D study. J Infect Dis. 2011 Aug 15;204(4):521-5. doi: 10.1093/infdis/jir329. PMID 21791653
- [Result] Pursuing Later Treatment Options II (PLATO II) project team; Collaboration of Observational HIV Epidemiological Research Europe (COHERE) Group; Nakagawa F, Lodwick R, Costagliola D, van Sighem A, Torti C, Podzamczer D, Mocroft A, Ledergerber B, Dorrucci M, Cozzi-Lepri A, Jansen K, Masquelier B, Garcia F, De Wit S, Stephan C, Obel N, Fatkenhaeuer G, Castagna A, Sambatakou H, Mussini C, Ghosn J, Zangerle R, Duval X, Meyer L, Perez-Hoyos S, Fabre Colin C, Kjaer J, Chene G, Grarup J, Phillips A. Calendar time trends in the incidence and prevalence of triple-class virologic failure in antiretroviral drug-experienced people with HIV in Europe. J Acquir Immune Defic Syndr. 2012 Mar 1;59(3):294-9. doi: 10.1097/QAI.0b013e31823fe66b. PMID 22083070
- [Result] Wittkop L, Gunthard HF, de Wolf F, Dunn D, Cozzi-Lepri A, de Luca A, Kucherer C, Obel N, von Wyl V, Masquelier B, Stephan C, Torti C, Antinori A, Garcia F, Judd A, Porter K, Thiebaut R, Castro H, van Sighem AI, Colin C, Kjaer J, Lundgren JD, Paredes R, Pozniak A, Clotet B, Phillips A, Pillay D, Chene G; EuroCoord-CHAIN study group. Effect of transmitted drug resistance on virological and immunological response to initial combination antiretroviral therapy for HIV (EuroCoord-CHAIN joint project): a European multicohort study. Lancet Infect Dis. 2011 May;11(5):363-71. doi: 10.1016/S1473-3099(11)70032-9. Epub 2011 Feb 25. PMID 21354861
- [Result] Reekie J, Mocroft A, Ledergerber B, Beniowski M, Clotet B, van Lunzen J, Chiesi A, Pradier C, Machala L, Lundgren JD; EuroSIDA Study Group. History of viral suppression on combination antiretroviral therapy as a predictor of virological failure after a treatment change. HIV Med. 2010 Aug;11(7):469-78. doi: 10.1111/j.1468-1293.2009.00816.x. Epub 2010 Feb 22. PMID 20201975
- [Result] Soriano V, Mocroft A, Peters L, Rockstroh J, Antunes F, Kirkby N, de Wit S, Monforte Ad, Flisiak R, Lundgren J; EuroSIDA. Predictors of hepatitis B virus genotype and viraemia in HIV-infected patients with chronic hepatitis B in Europe. J Antimicrob Chemother. 2010 Mar;65(3):548-55. doi: 10.1093/jac/dkp479. Epub 2010 Jan 5. PMID 20051475
- [Result] Pursuing Later Treatment Options II (PLATO II) Project Team for the Collaboration of Observational HIV Epidemiological Research Europe (COHERE); Lodwick R, Costagliola D, Reiss P, Torti C, Teira R, Dorrucci M, Ledergerber B, Mocroft A, Podzamczer D, Cozzi-Lepri A, Obel N, Masquelier B, Staszewski S, Garcia F, De Wit S, Castagna A, Antinori A, Judd A, Ghosn J, Touloumi G, Mussini C, Duval X, Ramos J, Meyer L, Warsawski J, Thorne C, Masip J, Perez-Hoyos S, Pillay D, van Sighem A, Lo Caputo S, Gunthard H, Paredes R, De Luca A, Paraskevis D, Fabre-Colin C, Kjaer J, Chene G, Lundgren JD, Phillips AN. Triple-class virologic failure in HIV-infected patients undergoing antiretroviral therapy for up to 10 years. Arch Intern Med. 2010 Mar 8;170(5):410-9. doi: 10.1001/archinternmed.2009.472. PMID 20212176
- [Result] Reekie J, Kosa C, Engsig F, Monforte Ad, Wiercinska-Drapalo A, Domingo P, Antunes F, Clumeck N, Kirk O, Lundgren JD, Mocroft A; EuroSIDA Study Group. Relationship between current level of immunodeficiency and non-acquired immunodeficiency syndrome-defining malignancies. Cancer. 2010 Nov 15;116(22):5306-15. doi: 10.1002/cncr.25311. PMID 20661911
- [Result] Mocroft A, Kirk O, Reiss P, De Wit S, Sedlacek D, Beniowski M, Gatell J, Phillips AN, Ledergerber B, Lundgren JD; EuroSIDA Study Group. Estimated glomerular filtration rate, chronic kidney disease and antiretroviral drug use in HIV-positive patients. AIDS. 2010 Jul 17;24(11):1667-78. doi: 10.1097/QAD.0b013e328339fe53. PMID 20523203
- [Result] Antiretroviral Therapy Cohort Collaboration. Causes of death in HIV-1-infected patients treated with antiretroviral therapy, 1996-2006: collaborative analysis of 13 HIV cohort studies. Clin Infect Dis. 2010 May 15;50(10):1387-96. doi: 10.1086/652283. PMID 20380565
- [Result] Opportunistic Infections Project Team of the Collaboration of Observational HIV Epidemiological Research in Europe (COHERE); Mocroft A, Reiss P, Kirk O, Mussini C, Girardi E, Morlat P, Stephan C, De Wit S, Doerholt K, Ghosn J, Bucher HC, Lundgren JD, Chene G, Miro JM, Furrer H. Is it safe to discontinue primary Pneumocystis jiroveci pneumonia prophylaxis in patients with virologically suppressed HIV infection and a CD4 cell count <200 cells/microL? Clin Infect Dis. 2010 Sep 1;51(5):611-9. doi: 10.1086/655761. PMID 20645862
- [Result] Mocroft A, Phillips AN, Ledergerber B, Smith C, Bogner JR, Lacombe K, Wiercinska-Drapalo A, Reiss P, Kirk O, Lundgren JD; EuroSIDA Study Group. Estimated average annual rate of change of CD4(+) T-cell counts in patients on combination antiretroviral therapy. Antivir Ther. 2010;15(4):563-70. doi: 10.3851/IMP1559. PMID 20587849
- [Result] Trullas JC, Mocroft A, Cofan F, Tourret J, Moreno A, Bagnis CI, Fux CA, Katlama C, Reiss P, Lundgren J, Gatell JM, Kirk O, Miro JM; EuroSIDA Investigators. Dialysis and renal transplantation in HIV-infected patients: a European survey. J Acquir Immune Defic Syndr. 2010 Dec 15;55(5):582-9. doi: 10.1097/QAI.0b013e3181efbe59. PMID 20811290
- [Result] Friis-Moller N, Thiebaut R, Reiss P, Weber R, Monforte AD, De Wit S, El-Sadr W, Fontas E, Worm S, Kirk O, Phillips A, Sabin CA, Lundgren JD, Law MG; DAD study group. Predicting the risk of cardiovascular disease in HIV-infected patients: the data collection on adverse effects of anti-HIV drugs study. Eur J Cardiovasc Prev Rehabil. 2010 Oct;17(5):491-501. doi: 10.1097/HJR.0b013e328336a150. PMID 20543702
- [Result] Worm SW, Friis-Moller N, Bruyand M, D'Arminio Monforte A, Rickenbach M, Reiss P, El-Sadr W, Phillips A, Lundgren J, Sabin C; D:A:D study group. High prevalence of the metabolic syndrome in HIV-infected patients: impact of different definitions of the metabolic syndrome. AIDS. 2010 Jan 28;24(3):427-35. doi: 10.1097/QAD.0b013e328334344e. PMID 19910787
- [Result] Worm SW, Sabin C, Weber R, Reiss P, El-Sadr W, Dabis F, De Wit S, Law M, Monforte AD, Friis-Moller N, Kirk O, Fontas E, Weller I, Phillips A, Lundgren J. Risk of myocardial infarction in patients with HIV infection exposed to specific individual antiretroviral drugs from the 3 major drug classes: the data collection on adverse events of anti-HIV drugs (D:A:D) study. J Infect Dis. 2010 Feb 1;201(3):318-30. doi: 10.1086/649897. PMID 20039804
- [Result] Data Collection on Adverse Events of Anti-HIV drugs (D:A:D) Study Group; Smith C, Sabin CA, Lundgren JD, Thiebaut R, Weber R, Law M, Monforte Ad, Kirk O, Friis-Moller N, Phillips A, Reiss P, El Sadr W, Pradier C, Worm SW. Factors associated with specific causes of death amongst HIV-positive individuals in the D:A:D Study. AIDS. 2010 Jun 19;24(10):1537-48. doi: 10.1097/QAD.0b013e32833a0918. PMID 20453631
- [Result] Data Collection on Adverse Events of Anti-HIV Drugs (D:A:D) Study Group; Weber R, Sabin C, Reiss P, de Wit S, Worm SW, Law M, Dabis F, D'Arminio Monforte A, Fontas E, El-Sadr W, Kirk O, Rickenbach M, Phillips A, Ledergerber B, Lundgren J. HBV or HCV coinfections and risk of myocardial infarction in HIV-infected individuals: the D:A:D Cohort Study. Antivir Ther. 2010;15(8):1077-86. doi: 10.3851/IMP1681. PMID 21149914
- [Result] Peters L, Mocroft A, Soriano V, Rockstroh JK, Losso M, Valerio L, Aldins P, Reiss P, Ledergerber B, Lundgren JD; EuroSIDA Study Group. Hepatitis C virus coinfection does not influence the CD4 cell recovery in HIV-1-infected patients with maximum virologic suppression. J Acquir Immune Defic Syndr. 2009 Apr 15;50(5):457-63. doi: 10.1097/qai.0b013e318198a0e1. PMID 19360931
- [Result] Cozzi-Lepri A, Phillips AN, Martinez-Picado J, Monforte Ad, Katlama C, Eg Hansen AB, Horban A, Bruun J, Clotet B, Lundgren JD; EuroSIDA Study Group. Rate of accumulation of thymidine analogue mutations in patients continuing to receive virologically failing regimens containing zidovudine or stavudine: implications for antiretroviral therapy programs in resource-limited settings. J Infect Dis. 2009 Sep 1;200(5):687-97. doi: 10.1086/604731. PMID 19604043
- [Result] Kesselring AM, Wit FW, Sabin CA, Lundgren JD, Gill MJ, Gatell JM, Rauch A, Montaner JS, de Wolf F, Reiss P, Mocroft A; Nevirapine Toxicity Multicohort Collaboration. Risk factors for treatment-limiting toxicities in patients starting nevirapine-containing antiretroviral therapy. AIDS. 2009 Aug 24;23(13):1689-99. doi: 10.1097/QAD.0b013e32832d3b54. PMID 19487907
- [Result] Worm SW, De Wit S, Weber R, Sabin CA, Reiss P, El-Sadr W, Monforte AD, Kirk O, Fontas E, Dabis F, Law MG, Lundgren JD, Friis-Moller N. Diabetes mellitus, preexisting coronary heart disease, and the risk of subsequent coronary heart disease events in patients infected with human immunodeficiency virus: the Data Collection on Adverse Events of Anti-HIV Drugs (D:A:D Study). Circulation. 2009 Feb 17;119(6):805-11. doi: 10.1161/CIRCULATIONAHA.108.790857. Epub 2009 Feb 2. PMID 19188509
- [Result] Worm SW, Sabin CA, Reiss P, El-Sadr W, Monforte Ad, Pradier C, Thiebaut R, Law M, Rickenbach M, De Wit S, Lundgren JD, Friis-Moller N. Presence of the metabolic syndrome is not a better predictor of cardiovascular disease than the sum of its components in HIV-infected individuals: data collection on adverse events of anti-HIV drugs (D:A:D) study. Diabetes Care. 2009 Mar;32(3):474-80. doi: 10.2337/dc08-1394. Epub 2008 Dec 3. PMID 19056612
- [Result] When To Start Consortium; Sterne JA, May M, Costagliola D, de Wolf F, Phillips AN, Harris R, Funk MJ, Geskus RB, Gill J, Dabis F, Miro JM, Justice AC, Ledergerber B, Fatkenheuer G, Hogg RS, Monforte AD, Saag M, Smith C, Staszewski S, Egger M, Cole SR. Timing of initiation of antiretroviral therapy in AIDS-free HIV-1-infected patients: a collaborative analysis of 18 HIV cohort studies. Lancet. 2009 Apr 18;373(9672):1352-63. doi: 10.1016/S0140-6736(09)60612-7. Epub 2009 Apr 8. PMID 19361855
- [Result] Collaboration of Observational HIV Epidemiological Research Europe (COHERE) study group; Bohlius J, Schmidlin K, Costagliola D, Fatkenheuer G, May M, Caro Murillo AM, Mocroft A, Bonnet F, Clifford G, Touloumi G, Miro JM, Chene G, Lundgren J, Egger M. Prognosis of HIV-associated non-Hodgkin lymphoma in patients starting combination antiretroviral therapy. AIDS. 2009 Sep 24;23(15):2029-37. doi: 10.1097/QAD.0b013e32832e531c. PMID 19531926
- [Result] Collaboration of Observational HIV Epidemiological Research Europe (COHERE) Study Group; Bohlius J, Schmidlin K, Costagliola D, Fatkenheuer G, May M, Caro-Murillo AM, Mocroft A, Bonnet F, Clifford G, Karafoulidou A, Miro JM, Lundgren J, Chene G, Egger M. Incidence and risk factors of HIV-related non-Hodgkin's lymphoma in the era of combination antiretroviral therapy: a European multicohort study. Antivir Ther. 2009;14(8):1065-74. doi: 10.3851/IMP1462. PMID 20032536
- [Result] Podlekareva DN, Mocroft A, Post FA, Riekstina V, Miro JM, Furrer H, Bruyand M, Panteleev AM, Rakhmanova AG, Girardi E, Losso MH, Toibaro JJ, Cayla J, Miller RF, Obel N, Skrahina A, Chentsova N, Lundgren JD, Kirk O; HIV/TB Study Writing Group. Mortality from HIV and TB coinfections is higher in Eastern Europe than in Western Europe and Argentina. AIDS. 2009 Nov 27;23(18):2485-95. doi: 10.1097/QAD.0b013e3283326879. PMID 19898216
- [Result] antiretroviral therapy cohort collaboration (ART-CC); Lanoy E, May M, Mocroft A, Phillip A, Justice A, Chene G, Furrer H, Sterling T, Monforte AD, Force L, Gill J, Harris R, Hogg RS, Rockstroh J, Saag M, Khaykin P, de Wolf F, Sterne JA, Costagliola D. Prognosis of patients treated with cART from 36 months after initiation, according to current and previous CD4 cell count and plasma HIV-1 RNA measurements. AIDS. 2009 Oct 23;23(16):2199-208. doi: 10.1097/QAD.0b013e3283305a00. PMID 19779320
- [Result] Moore DM, Harris R, Lima V, Hogg B, May M, Yip B, Justice A, Mocroft A, Reiss P, Lampe F, Chene G, Costagliola D, Elzi L, Mugavero MJ, Monforte AD, Sabin C, Podzamczer D, Fatkenheuer G, Staszewski S, Gill J, Sterne JA; Antiretroviral Therapy Cohort Collaboration. Effect of baseline CD4 cell counts on the clinical significance of short-term immunologic response to antiretroviral therapy in individuals with virologic suppression. J Acquir Immune Defic Syndr. 2009 Nov 1;52(3):357-63. doi: 10.1097/QAI.0b013e3181b62933. PMID 19668084
- [Result] Antiretroviral Therapy Cohort Collaboration (ART-CC); Mocroft A, Sterne JA, Egger M, May M, Grabar S, Furrer H, Sabin C, Fatkenheuer G, Justice A, Reiss P, d'Arminio Monforte A, Gill J, Hogg R, Bonnet F, Kitahata M, Staszewski S, Casabona J, Harris R, Saag M. Variable impact on mortality of AIDS-defining events diagnosed during combination antiretroviral therapy: not all AIDS-defining conditions are created equal. Clin Infect Dis. 2009 Apr 15;48(8):1138-51. doi: 10.1086/597468. PMID 19275498
- [Result] Mocroft A, Horban A, Clotet B, d'Arminio Monforte A, Bogner JR, Aldins P, Staub T, Antunes F, Katlama C, Lundgren JD; EuroSIDA Study Group. Regional differences in the risk of triple class failure in European patients starting combination antiretroviral therapy after 1 January 1999. HIV Med. 2008 Jan;9(1):41-6. doi: 10.1111/j.1468-1293.2008.00519.x. PMID 18199171
- [Result] Mocroft A, Kirk O, Aldins P, Chies A, Blaxhult A, Chentsova N, Vetter N, Dabis F, Gatell J, Lundgren JD; EuroSIDA study group. Loss to follow-up in an international, multicentre observational study. HIV Med. 2008 May;9(5):261-9. doi: 10.1111/j.1468-1293.2008.00557.x. PMID 18400074
- [Result] D:A:D Study Group; Sabin CA, Worm SW, Weber R, Reiss P, El-Sadr W, Dabis F, De Wit S, Law M, D'Arminio Monforte A, Friis-Moller N, Kirk O, Pradier C, Weller I, Phillips AN, Lundgren JD. Use of nucleoside reverse transcriptase inhibitors and risk of myocardial infarction in HIV-infected patients enrolled in the D:A:D study: a multi-cohort collaboration. Lancet. 2008 Apr 26;371(9622):1417-26. doi: 10.1016/S0140-6736(08)60423-7. Epub 2008 Apr 2. PMID 18387667
- [Result] Deforche K, Cozzi-Lepri A, Theys K, Clotet B, Camacho RJ, Kjaer J, Van Laethem K, Phillips A, Moreau Y, Lundgren JD, Vandamme AM; EuroSIDA Study Group. Modelled in vivo HIV fitness under drug selective pressure and estimated genetic barrier towards resistance are predictive for virological response. Antivir Ther. 2008;13(3):399-407. PMID 18572753
- [Result] Podlekareva D, Mocroft A, Kirk O, Reiss P, Aldins P, Katlama C, Kovari H, Stellbrink HJ, D'Arminio Monforte A, Lundgren JD; Eurosida Study Group. Fungal infection as a risk factor for HIV disease progression among patients with a CD4 count above 200/microl in the era of cART. Scand J Infect Dis. 2008;40(11-12):908-13. doi: 10.1080/00365540802227094. PMID 18609197
- [Result] Cozzi-Lepri A, Phillips AN, Clotet B, Mocroft A, Ruiz L, Kirk O, Lazzarin A, Wiercinska-Drapalo A, Karlsson A, Lundgren JD; EuroSIDA Study Group. Detection of HIV drug resistance during antiretroviral treatment and clinical progression in a large European cohort study. AIDS. 2008 Oct 18;22(16):2187-98. doi: 10.1097/QAD.0b013e328310e04f. PMID 18832882
- [Result] Reekie J, Mocroft A, Sambatakou H, Machala L, Chiesi A, van Lunzen J, Clumeck N, Kirk O, Gazzard B, Lundgren JD; EuroSIDA Study Group. Does less frequent routine monitoring of patients on a stable, fully suppressed cART regimen lead to an increased risk of treatment failure? AIDS. 2008 Nov 12;22(17):2381-90. doi: 10.1097/QAD.0b013e328317a6eb. PMID 18981778
- [Result] Soriano V, Mocroft A, Rockstroh J, Ledergerber B, Knysz B, Chaplinskas S, Peters L, Karlsson A, Katlama C, Toro C, Kupfer B, Vogel M, Lundgren J; EuroSIDA Study Group. Spontaneous viral clearance, viral load, and genotype distribution of hepatitis C virus (HCV) in HIV-infected patients with anti-HCV antibodies in Europe. J Infect Dis. 2008 Nov 1;198(9):1337-44. doi: 10.1086/592171. PMID 18767985
- [Result] Antiretroviral Therapy Cohort Collaboration (ART-CC); Mugavero MJ, May M, Harris R, Saag MS, Costagliola D, Egger M, Phillips A, Gunthard HF, Dabis F, Hogg R, de Wolf F, Fatkenheuer G, Gill MJ, Justice A, D'Arminio Monforte A, Lampe F, Miro JM, Staszewski S, Sterne JA. Does short-term virologic failure translate to clinical events in antiretroviral-naive patients initiating antiretroviral therapy in clinical practice? AIDS. 2008 Nov 30;22(18):2481-92. doi: 10.1097/QAD.0b013e328318f130. PMID 19005271
- [Result] Antiretroviral Therapy Cohort Collaboration. Life expectancy of individuals on combination antiretroviral therapy in high-income countries: a collaborative analysis of 14 cohort studies. Lancet. 2008 Jul 26;372(9635):293-9. doi: 10.1016/S0140-6736(08)61113-7. PMID 18657708
- [Result] Monforte Ad, Abrams D, Pradier C, Weber R, Reiss P, Bonnet F, Kirk O, Law M, De Wit S, Friis-Moller N, Phillips AN, Sabin CA, Lundgren JD; Data Collection on Adverse Events of Anti-HIV Drugs (D:A:D) Study Group. HIV-induced immunodeficiency and mortality from AIDS-defining and non-AIDS-defining malignancies. AIDS. 2008 Oct 18;22(16):2143-53. doi: 10.1097/QAD.0b013e3283112b77. PMID 18832878
- [Result] Data Collection on Adverse Events of Anti-HIV Drugs Study Group; Sabin CA, d'Arminio Monforte A, Friis-Moller N, Weber R, El-Sadr WM, Reiss P, Kirk O, Mercie P, Law MG, De Wit S, Pradier C, Phillips AN, Lundgren JD. Changes over time in risk factors for cardiovascular disease and use of lipid-lowering drugs in HIV-infected individuals and impact on myocardial infarction. Clin Infect Dis. 2008 Apr 1;46(7):1101-10. doi: 10.1086/528862. PMID 18461712
- [Result] Collaboration of Observational HIV Epidemiological Research Europe (COHERE) Study Group; Sabin CA, Smith CJ, d'Arminio Monforte A, Battegay M, Gabiano C, Galli L, Geelen S, Gibb D, Guiguet M, Judd A, Leport C, Dabis F, Pantazis N, Porter K, Raffi F, Thorne C, Torti C, Walker S, Warszawski J, Wintergerst U, Chene G, Lundgren J. Response to combination antiretroviral therapy: variation by age. AIDS. 2008 Jul 31;22(12):1463-73. doi: 10.1097/QAD.0b013e3282f88d02. PMID 18614870
- [Result] Harris RJ, Sterne JA, Abgrall S, Dabis F, Reiss P, Saag M, Phillips AN, Chene G, Gill JM, Justice AC, Rockstroh J, Sabin CA, Mocroft A, Bucher HC, Hogg RS, Monforte AD, May M, Egger M; Antiretroviral Therapy Cohort Collaboration. Prognostic importance of anaemia in HIV type-1-infected patients starting antiretroviral therapy: collaborative analysis of prospective cohort studies. Antivir Ther. 2008;13(8):959-67. PMID 19195321
- [Result] De Wit S, Sabin CA, Weber R, Worm SW, Reiss P, Cazanave C, El-Sadr W, Monforte Ad, Fontas E, Law MG, Friis-Moller N, Phillips A; Data Collection on Adverse Events of Anti-HIV Drugs (D:A:D) study. Incidence and risk factors for new-onset diabetes in HIV-infected patients: the Data Collection on Adverse Events of Anti-HIV Drugs (D:A:D) study. Diabetes Care. 2008 Jun;31(6):1224-9. doi: 10.2337/dc07-2013. Epub 2008 Feb 11. PMID 18268071
- [Result] Strategies for Management of Anti-Retroviral Therapy/INSIGHT; DAD Study Groups. Use of nucleoside reverse transcriptase inhibitors and risk of myocardial infarction in HIV-infected patients. AIDS. 2008 Sep 12;22(14):F17-24. doi: 10.1097/QAD.0b013e32830fe35e. PMID 18753925
- [Result] Cozzi-Lepri A, Phillips AN, Ruiz L, Clotet B, Loveday C, Kjaer J, Mens H, Clumeck N, Viksna L, Antunes F, Machala L, Lundgren JD; EuroSIDA Study Group. Evolution of drug resistance in HIV-infected patients remaining on a virologically failing combination antiretroviral therapy regimen. AIDS. 2007 Mar 30;21(6):721-32. doi: 10.1097/QAD.0b013e3280141fdf. PMID 17413693
- [Result] Holkmann Olsen C, Mocroft A, Kirk O, Vella S, Blaxhult A, Clumeck N, Fisher M, Katlama C, Phillips AN, Lundgren JD; EuroSIDA study group. Interruption of combination antiretroviral therapy and risk of clinical disease progression to AIDS or death. HIV Med. 2007 Mar;8(2):96-104. doi: 10.1111/j.1468-1293.2007.00436.x. PMID 17352766
- [Result] DAD Study Group; Friis-Moller N, Reiss P, Sabin CA, Weber R, Monforte Ad, El-Sadr W, Thiebaut R, De Wit S, Kirk O, Fontas E, Law MG, Phillips A, Lundgren JD. Class of antiretroviral drugs and the risk of myocardial infarction. N Engl J Med. 2007 Apr 26;356(17):1723-35. doi: 10.1056/NEJMoa062744. PMID 17460226
- [Result] Mocroft A, Kirk O, Gatell J, Reiss P, Gargalianos P, Zilmer K, Beniowski M, Viard JP, Staszewski S, Lundgren JD. Chronic renal failure among HIV-1-infected patients. AIDS. 2007 May 31;21(9):1119-27. doi: 10.1097/QAD.0b013e3280f774ee. PMID 17502722
- [Result] Mocroft A, Phillips AN, Gatell J, Ledergerber B, Fisher M, Clumeck N, Losso M, Lazzarin A, Fatkenheuer G, Lundgren JD; EuroSIDA study group. Normalisation of CD4 counts in patients with HIV-1 infection and maximum virological suppression who are taking combination antiretroviral therapy: an observational cohort study. Lancet. 2007 Aug 4;370(9585):407-13. doi: 10.1016/S0140-6736(07)60948-9. PMID 17659333
- [Result] Kowalska JD, Mocroft A, Blaxhult A, Colebunders R, van Lunzen J, Podlekareva D, Hansen AB, Machala L, Yust I, Benfield T; EuroSIDA Study Group. Current hemoglobin levels are more predictive of disease progression than hemoglobin measured at baseline in patients receiving antiretroviral treatment for HIV type 1 infection. AIDS Res Hum Retroviruses. 2007 Oct;23(10):1183-8. doi: 10.1089/aid.2006.0292. PMID 17961102
- [Result] Ceccherini-Silberstein F, Cozzi-Lepri A, Ruiz L, Mocroft A, Phillips AN, Olsen CH, Gatell JM, Gunthard HF, Reiss P, Perno CF, Clotet B, Lundgren JD; EuroSIDA Study Group. Impact of HIV-1 reverse transcriptase polymorphism F214L on virological response to thymidine analogue-based regimens in antiretroviral therapy (ART)-naive and ART-experienced patients. J Infect Dis. 2007 Oct 15;196(8):1180-90. doi: 10.1086/521678. Epub 2007 Sep 19. PMID 17955437
- [Result] Fox ZV, Geretti AM, Kjaer J, Dragsted UB, Phillips AN, Gerstoft J, Staszewski S, Clotet B, von Wyl V, Lundgren JD. The ability of four genotypic interpretation systems to predict virological response to ritonavir-boosted protease inhibitors. AIDS. 2007 Oct 1;21(15):2033-42. doi: 10.1097/QAD.0b013e32825a69e4. PMID 17885293
- [Result] Mocroft A, Staszewski S, Weber R, Gatell J, Rockstroh J, Gasiorowski J, Panos G, Monforte Ad, Rakhmanova A, Phillips AN, Lundgren JD; EuroSIDA study group. Risk of discontinuation of nevirapine due to toxicities in antiretroviral-naive and -experienced HIV-infected patients with high and low CD4+ T-cell counts. Antivir Ther. 2007;12(3):325-33. PMID 17591022
- [Result] Antiretroviral Therapy in Low-Income Countries Collaboration of the International epidemiological Databases to Evaluate AIDS (IeDEA); ART Cohort Collaboration; Brinkhof MW, Egger M, Boulle A, May M, Hosseinipour M, Sprinz E, Braitstein P, Dabis F, Reiss P, Bangsberg DR, Rickenbach M, Miro JM, Myer L, Mocroft A, Nash D, Keiser O, Pascoe M, van der Borght S, Schechter M. Tuberculosis after initiation of antiretroviral therapy in low-income and high-income countries. Clin Infect Dis. 2007 Dec 1;45(11):1518-21. doi: 10.1086/522986. Epub 2007 Oct 22. PMID 17990236
- [Result] Antiretroviral Therapy Cohort Collaboration. Importance of baseline prognostic factors with increasing time since initiation of highly active antiretroviral therapy: collaborative analysis of cohorts of HIV-1-infected patients. J Acquir Immune Defic Syndr. 2007 Dec 15;46(5):607-15. doi: 10.1097/QAI.0b013e31815b7dba. PMID 18043315
- [Result] May M, Sterne JA, Shipley M, Brunner E, d'Agostino R, Whincup P, Ben-Shlomo Y, Carr A, Ledergerber B, Lundgren JD, Phillips AN, Massaro J, Egger M. A coronary heart disease risk model for predicting the effect of potent antiretroviral therapy in HIV-1 infected men. Int J Epidemiol. 2007 Dec;36(6):1309-18. doi: 10.1093/ije/dym135. Epub 2007 Jul 25. PMID 17652317
- [Result] Sterne JA, May M, Bucher HC, Ledergerber B, Furrer H, Cavassini M, Bernasconi E, Hirschel B, Egger M; Swiss HIV Cohort. HAART and the heart: changes in coronary risk factors and implications for coronary risk in men starting antiretroviral therapy. J Intern Med. 2007 Mar;261(3):255-67. doi: 10.1111/j.1365-2796.2006.01761.x. PMID 17305648
- [Result] Llibre JM, Cozzi-Lepri A, La Rosa JA, Pedersen C, Ristola M, Losso M, Mocroft A, Mitsura VM, Ormaasen V, Maltez F, Beniowski M, Paredes R; Eurosida in Eurocoord. Long term effectiveness of once-daily unboosted atazanavir plus abacavir/lamivudine as a switch strategy in subjects with virological suppression. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19810. doi: 10.7448/IAS.17.4.19810. eCollection 2014. PMID 25397554
- [Result] Schultze A, Paredes R, Sabin C, Phillips AN, Pillay D, Kirk O, Lundgren JD, Pozniak A, Nelson M, Cozzi-Lepri A; Eurosida in Eurocoord. Detection of resistance mutations and CD4 slopes in individuals experiencing sustained virological failure. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19737. doi: 10.7448/IAS.17.4.19737. eCollection 2014. PMID 25397482
- [Result] Fontdevila MC, Cozzi-Lepri A, Phillips A, Julian MN, Bickel M, Sedlacek D, Kronborg G, Lazzarin A, Zilmer K, Clotet B, Lundgren JD, Paredes R. Plasma HIV-1 tropism and risk of short-term clinical progression to AIDS or death. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19685. doi: 10.7448/IAS.17.4.19685. eCollection 2014. PMID 25397435
- [Result] Mocroft A, Reiss P, Gasiorowski J, Ledergerber B, Kowalska J, Chiesi A, Gatell J, Rakhmanova A, Johnson M, Kirk O, Lundgren J; EuroSIDA Study Group. Serious fatal and nonfatal non-AIDS-defining illnesses in Europe. J Acquir Immune Defic Syndr. 2010 Oct;55(2):262-70. doi: 10.1097/QAI.0b013e3181e9be6b. PMID 20700060
- [Result] Young J, Bucher HC, Guenthard HF, Rickenbach M, Fux CA, Hirschel B, Cavassini M, Vernazza P, Bernasconi E, Battegay M; Swiss HIV Cohort Study. Virological and immunological responses to efavirenz or boosted lopinavir as first-line therapy for patients with HIV. Antivir Ther. 2009;14(6):771-9. doi: 10.3851/IMP1291. PMID 19812439
- [Result] Smith CJ, Mocroft A, Lundgren JD; EuroSIDA Study Group. Incidence of pancreatitis in HIV-infected patients, and the association with antiretroviral therapy. AIDS. 2008 May 11;22(8):997-8. doi: 10.1097/QAD.0b013e3282ffb0fd. No abstract available. PMID 18453864
- [Result] Bannister WP, Ruiz L, Loveday C, Vella S, Zilmer K, Kjaer J, Knysz B, Phillips AN, Mocroft A; EuroSIDA Study Group. HIV-1 subtypes and response to combination antiretroviral therapy in Europe. Antivir Ther. 2006;11(6):707-15. PMID 17310815
- [Result] Mocroft, Horban, Clumeck, Stellbrink, Monforte dA, Zilmer, Kirk, Gatell, Phillips, Lundgren; EuroSIDA Study Group. Comparison of single and boosted protease inhibitor versus nonnucleoside reverse transcriptase inhibitor-containing cART regimens in antiretroviral-naive patients starting cART after January 1, 2000. HIV Clin Trials. 2006 Nov-Dec;7(6):271-84. doi: 10.1310/hct0706-271. PMID 17208897
- [Result] Mocroft A, Rockstroh J, Soriano V, Kirk O, Viard JP, Caplinskas S, Gasiorowski J, Chiesi A, Phillips AN, Lundgren JD; EuroSIDA Study Group. Limited but increasing use of treatment for hepatitis C across Europe in patients coinfected with HIV and hepatitis C. Scand J Infect Dis. 2006;38(11-12):1092-7. doi: 10.1080/00365540600786515. PMID 17148084
- [Result] Mocroft A, Neaton J, Bebchuk J, Staszewski S, Antunes F, Knysz B, Law M, Phillips AN, Lundgren JD; EuroSIDA Study Group; ESPRIT Study Group. The feasibility of clinical endpoint trials in HIV infection in the highly active antiretroviral treatment (HAART) era. Clin Trials. 2006;3(2):119-32. doi: 10.1191/1740774506cn138oa. PMID 16773954
- [Result] Bannister WP, Kirk O, Gatell JM, Knysz B, Viard JP, Mens H, Monforte AD, Phillips AN, Mocroft A, Lundgren JD; EuroSIDA Study Group. Regional changes over time in initial virologic response rates to combination antiretroviral therapy across Europe. J Acquir Immune Defic Syndr. 2006 Jun;42(2):229-37. doi: 10.1097/01.qai.0000214815.95786.31. PMID 16760800
- [Result] Rockstroh JK. Influence of viral hepatitis on HIV infection. J Hepatol. 2006;44(1 Suppl):S25-7. doi: 10.1016/j.jhep.2005.11.007. Epub 2005 Nov 21. PMID 16338020
- [Result] Braitstein P, Brinkhof MW, Dabis F, Schechter M, Boulle A, Miotti P, Wood R, Laurent C, Sprinz E, Seyler C, Bangsberg DR, Balestre E, Sterne JA, May M, Egger M; Antiretroviral Therapy in Lower Income Countries (ART-LINC) Collaboration; ART Cohort Collaboration (ART-CC) groups. Mortality of HIV-1-infected patients in the first year of antiretroviral therapy: comparison between low-income and high-income countries. Lancet. 2006 Mar 11;367(9513):817-24. doi: 10.1016/S0140-6736(06)68337-2. PMID 16530575
- [Result] Law MG, Friis-Moller N, El-Sadr WM, Weber R, Reiss P, D'Arminio Monforte A, Thiebaut R, Morfeldt L, De Wit S, Pradier C, Calvo G, Kirk O, Sabin CA, Phillips AN, Lundgren JD; D:A:D Study Group. The use of the Framingham equation to predict myocardial infarctions in HIV-infected patients: comparison with observed events in the D:A:D Study. HIV Med. 2006 May;7(4):218-30. doi: 10.1111/j.1468-1293.2006.00362.x. PMID 16630034
- [Result] Mocroft A, Phillips AN, Ledergerber B, Katlama C, Chiesi A, Goebel FD, Knysz B, Antunes F, Reiss P, Lundgren JD. Relationship between antiretrovirals used as part of a cART regimen and CD4 cell count increases in patients with suppressed viremia. AIDS. 2006 May 12;20(8):1141-50. doi: 10.1097/01.aids.0000226954.95094.39. PMID 16691065
- [Result] Weber R, Sabin CA, Friis-Moller N, Reiss P, El-Sadr WM, Kirk O, Dabis F, Law MG, Pradier C, De Wit S, Akerlund B, Calvo G, Monforte Ad, Rickenbach M, Ledergerber B, Phillips AN, Lundgren JD. Liver-related deaths in persons infected with the human immunodeficiency virus: the D:A:D study. Arch Intern Med. 2006 Aug 14-28;166(15):1632-41. doi: 10.1001/archinte.166.15.1632. PMID 16908797
- [Result] Puoti M, Cozzi-Lepri A, Paraninfo G, Arici C, Moller NF, Lundgren JD, Ledergerber B, Rickenbach M, Suarez-Lozano I, Garrido M, Dabis F, Winnock M, Milazzo L, Gervais A, Raffi F, Gill J, Rockstroh J, Ourishi N, Mussini C, Castagna A, De Luca A, Monforte Ad; HBV-HIV International Intercohort Study Group. Impact of lamivudine on the risk of liver-related death in 2,041 HBsAg- and HIV-positive individuals: results from an inter-cohort analysis. Antivir Ther. 2006;11(5):567-74. doi: 10.1177/135965350601100509. PMID 16964824
- [Result] May MT, Sterne JA, Costagliola D, Sabin CA, Phillips AN, Justice AC, Dabis F, Gill J, Lundgren J, Hogg RS, de Wolf F, Fatkenheuer G, Staszewski S, d'Arminio Monforte A, Egger M; Antiretroviral Therapy (ART) Cohort Collaboration. HIV treatment response and prognosis in Europe and North America in the first decade of highly active antiretroviral therapy: a collaborative analysis. Lancet. 2006 Aug 5;368(9534):451-8. doi: 10.1016/S0140-6736(06)69152-6. PMID 16890831
- [Result] Antiretroviral Therapy Cohort Collaboration. Rates of disease progression according to initial highly active antiretroviral therapy regimen: a collaborative analysis of 12 prospective cohort studies. J Infect Dis. 2006 Sep 1;194(5):612-22. doi: 10.1086/506362. Epub 2006 Jul 31. PMID 16897660
- [Result] Cozzi-Lepri A, Ruiz L, Loveday C, Phillips AN, Clotet B, Reiss P, Ledergerber B, Holkmann C, Staszewski S, Lundgren JD; EuroSIDA Study Group. Thymidine analogue mutation profiles: factors associated with acquiring specific profiles and their impact on the virological response to therapy. Antivir Ther. 2005;10(7):791-802. PMID 16312176
- [Result] Mocroft A, Rockstroh J, Soriano V, Ledergerber B, Kirk O, Vinogradova E, Reiss P, Katlama C, Phillips AN, Lundgren JD; EuroSIDA Study Group. Are specific antiretrovirals associated with an increased risk of discontinuation due to toxicities or patient/physician choice in patients with hepatitis C virus coinfection? Antivir Ther. 2005;10(7):779-90. PMID 16312175
- [Result] Mocroft A, Soriano V, Rockstroh J, Reiss P, Kirk O, de Wit S, Gatell J, Clotet B, Phillips AN, Lundgren JD; EuroSIDA Study Group. Is there evidence for an increase in the death rate from liver-related disease in patients with HIV? AIDS. 2005 Dec 2;19(18):2117-25. doi: 10.1097/01.aids.0000194799.43799.ea. PMID 16284461
- [Result] Mocroft A, Phillips AN, Soriano V, Rockstroh J, Blaxhult A, Katlama C, Boron-Kaczmarska A, Viksna L, Kirk O, Lundgren JD; EuroSIDA Study Group. Reasons for stopping antiretrovirals used in an initial highly active antiretroviral regimen: increased incidence of stopping due to toxicity or patient/physician choice in patients with hepatitis C coinfection. AIDS Res Hum Retroviruses. 2005 Sep;21(9):743-52. doi: 10.1089/aid.2005.21.743. PMID 16218797
- [Result] Rockstroh JK, Mocroft A, Soriano V, Tural C, Losso MH, Horban A, Kirk O, Phillips A, Ledergerber B, Lundgren J; EuroSIDA Study Group. Influence of hepatitis C virus infection on HIV-1 disease progression and response to highly active antiretroviral therapy. J Infect Dis. 2005 Sep 15;192(6):992-1002. doi: 10.1086/432762. Epub 2005 Aug 11. PMID 16107951
- [Result] Mocroft A, Phillips AN, Soriano V, Rockstroh J, Blaxhult A, Katlama C, Boron-Kaczmarska A, Viksna L, Kirk O, Lundgren JD; EuroSIDA Study Group. Reasons for stopping antiretrovirals used in an initial highly active antiretroviral regimen: increased incidence of stopping due to toxicity or patient/physician choice in patients with hepatitis C coinfection. AIDS Res Hum Retroviruses. 2005 Jun;21(6):527-36. doi: 10.1089/aid.2005.21.527. PMID 15989457
- [Result] Mocroft A, Oancea C, van Lunzen J, Vanhems P, Banhegyi D, Chiesi A, Vinogradova E, Maayan S, Phillips AN, Lundgren J; EuroSIDA study group. Decline in esophageal candidiasis and use of antimycotics in European patients with HIV. Am J Gastroenterol. 2005 Jul;100(7):1446-54. doi: 10.1111/j.1572-0241.2005.41949.x. PMID 15984964
- [Result] Olsen CH, Gatell J, Ledergerber B, Katlama C, Friis-Moller N, Weber J, Horban A, Staszewski S, Lundgren JD, Phillips AN; EuroSIDA Study Group. Risk of AIDS and death at given HIV-RNA and CD4 cell count, in relation to specific antiretroviral drugs in the regimen. AIDS. 2005 Feb 18;19(3):319-30. PMID 15718843
- [Result] Mocroft A, Gatell J, Reiss P, Ledergerber B, Kirk O, Vella S, Blaxhult A, Phillips AN, Lundgren J; EuroSIDA study group. Causes of death in HIV infection: the key determinant to define the clinical response to anti-HIV therapy. AIDS. 2004 Nov 19;18(17):2333-7. doi: 10.1097/00002030-200411190-00018. PMID 15577550
- [Result] Phillips AN, Ledergerber B, Horban A, Reiss P, Chiesi A, Kirk O, Mulchany F, Fisher M, Machala L, Lundgren JD; EuroSIDA Study Group. Rate of viral rebound according to specific drugs in the regimen in 2120 patients with HIV suppression. AIDS. 2004 Sep 3;18(13):1795-804. doi: 10.1097/00002030-200409030-00008. PMID 15316340
- [Result] Lundgren JD, Mocroft A. Anemia and survival in human immunodeficiency virus. Clin Infect Dis. 2003;37 Suppl 4:S297-303. doi: 10.1086/376909. PMID 14581998
- [Result] Mocroft A, Ruiz L, Reiss P, Ledergerber B, Katlama C, Lazzarin A, Goebel FD, Phillips AN, Clotet B, Lundgren JD; EuroSIDA study group. Virological rebound after suppression on highly active antiretroviral therapy. AIDS. 2003 Aug 15;17(12):1741-51. doi: 10.1097/00002030-200308150-00003. PMID 12891060
- [Result] Cozzi-Lepri A, Phillips AN, Miller V, Katlama C, Ledergerber B, Vella S, Weber J, Bruun JN, Kirk O, Clotet B, Lundgrens JD. Changes in viral load in people with virological failure who remain on the same HAART regimen. Antivir Ther. 2003 Apr;8(2):127-36. PMID 12741625
- [Result] Moore AL, Kirk O, Johnson AM, Katlama C, Blaxhult A, Dietrich M, Colebunders R, Chiesi A, Lungren JD, Phillips AN; EuroSIDA group. Virologic, immunologic, and clinical response to highly active antiretroviral therapy: the gender issue revisited. J Acquir Immune Defic Syndr. 2003 Apr 1;32(4):452-61. doi: 10.1097/00126334-200304010-00017. PMID 12640206
- [Result] Blaxhult A, Fox Z, Colebunders R, Francioli P, Ben-Ishai Z, Fatkenheuer G, Parkin JM, Vanhems P, Phillips AN, Kirk O; EuroSIDA Study Group. Regional and temporal changes in AIDS in Europe before HAART. Epidemiol Infect. 2002 Dec;129(3):565-76. doi: 10.1017/s0950268802007719. PMID 12558340
- [Result] Kirk O, Pedersen C, Law M, Gulick RM, Moyle G, Montaner J, Eron JJ Jr, Phillips AN, Lundgren JD. Analysis of virological efficacy in trials of antiretroviral regimens: drawbacks of not including viral load measurements after premature discontinuation of therapy. Antivir Ther. 2002 Dec;7(4):271-81. PMID 12553482
- [Result] Kirk O, Reiss P, Uberti-Foppa C, Bickel M, Gerstoft J, Pradier C, Wit FW, Ledergerber B, Lundgren JD, Furrer H; European HIV Cohorts. Safe interruption of maintenance therapy against previous infection with four common HIV-associated opportunistic pathogens during potent antiretroviral therapy. Ann Intern Med. 2002 Aug 20;137(4):239-50. doi: 10.7326/0003-4819-137-4-200208200-00008. PMID 12186514
- [Result] Phillips AN, Pradier C, Lazzarin A, Clotet B, Goebel FD, Hermans P, Antunes F, Ledergerber B, Kirk O, Lundgren JD; EuroSIDA Study Group. Viral load outcome of non-nucleoside reverse transcriptase inhibitor regimens for 2203 mainly antiretroviral-experienced patients. AIDS. 2001 Dec 7;15(18):2385-95. doi: 10.1097/00002030-200112070-00006. PMID 11740189
- [Result] Phillips AN, Staszewski S, Weber R, Kirk O, Francioli P, Miller V, Vernazza P, Lundgren JD, Ledergerber B; Swiss HIV Cohort Study; Frakfurt HIV Clinic Cohort; EuroSIDA Study Group. HIV viral load response to antiretroviral therapy according to the baseline CD4 cell count and viral load. JAMA. 2001 Nov 28;286(20):2560-7. doi: 10.1001/jama.286.20.2560. PMID 11722270
- [Result] Kirk O, Pedersen C, Cozzi-Lepri A, Antunes F, Miller V, Gatell JM, Katlama C, Lazzarin A, Skinhoj P, Barton SE; EuroSIDA Study Group. Non-Hodgkin lymphoma in HIV-infected patients in the era of highly active antiretroviral therapy. Blood. 2001 Dec 1;98(12):3406-12. doi: 10.1182/blood.v98.12.3406. PMID 11719381
- [Result] Kirk O, Mocroft A, Pradier C, Bruun JN, Hemmer R, Clotet B, Miller V, Viard JP, Phillips AN, Lundgren JD; EuroSIDA Study Group. Clinical outcome among HIV-infected patients starting saquinavir hard gel compared to ritonavir or indinavir. AIDS. 2001 May 25;15(8):999-1008. doi: 10.1097/00002030-200105250-00008. PMID 11399982
- [Result] Norton M. Stopping PCP prophylaxis after suppressing HIV. GMHC Treat Issues. 1999 Apr;13(4):4-5. PMID 11366976
- [Result] Thiebaut R, El-Sadr WM, Friis-Moller N, Rickenbach M, Reiss P, Monforte AD, Morfeldt L, Fontas E, Kirk O, De Wit S, Calvo G, Law MG, Dabis F, Sabin CA, Lundgren JD; Data Collection of Adverse events of anti-HIV Drugs Study Group. Predictors of hypertension and changes of blood pressure in HIV-infected patients. Antivir Ther. 2005;10(7):811-23. doi: 10.1177/135965350501000706. PMID 16315369
- [Result] Girardi E, Sabin CA, d'Arminio Monforte A, Hogg B, Phillips AN, Gill MJ, Dabis F, Reiss P, Kirk O, Bernasconi E, Grabar S, Justice A, Staszewski S, Fatkenheuer G, Sterne JA; Antiretroviral Therapy Cohort Collaboration. Incidence of Tuberculosis among HIV-infected patients receiving highly active antiretroviral therapy in Europe and North America. Clin Infect Dis. 2005 Dec 15;41(12):1772-82. doi: 10.1086/498315. Epub 2005 Nov 11. PMID 16288403
- [Result] Sabine C; Antiretroviral Therapy (ART) Cohort Collaboration. AIDS events among individuals initiating HAART: do some patients experience a greater benefit from HAART than others? AIDS. 2005 Nov 18;19(17):1995-2000. doi: 10.1097/01.aids.0000189858.59559.d2. PMID 16260906
- [Result] May M, Porter K, Sterne JA, Royston P, Egger M. Prognostic model for HIV-1 disease progression in patients starting antiretroviral therapy was validated using independent data. J Clin Epidemiol. 2005 Oct;58(10):1033-41. doi: 10.1016/j.jclinepi.2005.02.015. PMID 16168349
- [Result] d'Arminio Monforte A, Sabin CA, Phillips A, Sterne J, May M, Justice A, Dabis F, Grabar S, Ledergerber B, Gill J, Reiss P, Egger M; Antiretroviral Therapy Cohort Collaboration. The changing incidence of AIDS events in patients receiving highly active antiretroviral therapy. Arch Intern Med. 2005 Feb 28;165(4):416-23. doi: 10.1001/archinte.165.4.416. PMID 15738371
- [Result] Fontas E, van Leth F, Sabin CA, Friis-Moller N, Rickenbach M, d'Arminio Monforte A, Kirk O, Dupon M, Morfeldt L, Mateu S, Petoumenos K, El-Sadr W, de Wit S, Lundgren JD, Pradier C, Reiss P; D:A:D Study Group. Lipid profiles in HIV-infected patients receiving combination antiretroviral therapy: are different antiretroviral drugs associated with different lipid profiles? J Infect Dis. 2004 Mar 15;189(6):1056-74. doi: 10.1086/381783. Epub 2004 Mar 2. PMID 14999610
- [Result] Ledergerber B, Lundgren JD, Walker AS, Sabin C, Justice A, Reiss P, Mussini C, Wit F, d'Arminio Monforte A, Weber R, Fusco G, Staszewski S, Law M, Hogg R, Lampe F, Gill MJ, Castelli F, Phillips AN; PLATO Collaboration. Predictors of trend in CD4-positive T-cell count and mortality among HIV-1-infected individuals with virological failure to all three antiretroviral-drug classes. Lancet. 2004 Jul 3-9;364(9428):51-62. doi: 10.1016/S0140-6736(04)16589-6. PMID 15234856
- [Result] d'Arminio A, Sabin CA, Phillips AN, Reiss P, Weber R, Kirk O, El-Sadr W, De Wit S, Mateu S, Petoumenos K, Dabis F, Pradier C, Morfeldt L, Lundgren JD, Friis-Moller N; Writing Committee of the D:A:D: Study Group. Cardio- and cerebrovascular events in HIV-infected persons. AIDS. 2004 Sep 3;18(13):1811-7. doi: 10.1097/00002030-200409030-00010. PMID 15316342
- [Result] Collaboration of HIV Cohorts. Nucleoside analogue use before and during highly active antiretroviral therapy and virus load rebound. J Infect Dis. 2004 Aug 15;190(4):675-87. doi: 10.1086/421707. Epub 2004 Jul 19. PMID 15272393
- [Result] Law M, Friis-Moller N, Weber R, Reiss P, Thiebaut R, Kirk O, d'Arminio Monforte A, Pradier C, Morfeldt L, Calvo G, El-Sadr W, De Wit S, Sabin CA, Lundgren JD; DAD Study Group. Modelling the 3-year risk of myocardial infarction among participants in the Data Collection on Adverse Events of Anti-HIV Drugs (DAD) study. HIV Med. 2003 Jan;4(1):1-10. doi: 10.1046/j.1468-1293.2003.00138.x. PMID 12534953
- [Result] May M, Royston P, Egger M, Justice AC, Sterne JA; ART Cohort Collaboration. Development and validation of a prognostic model for survival time data: application to prognosis of HIV positive patients treated with antiretroviral therapy. Stat Med. 2004 Aug 15;23(15):2375-98. doi: 10.1002/sim.1825. PMID 15273954
- [Result] Friis-Moller N, Weber R, Reiss P, Thiebaut R, Kirk O, d'Arminio Monforte A, Pradier C, Morfeldt L, Mateu S, Law M, El-Sadr W, De Wit S, Sabin CA, Phillips AN, Lundgren JD; DAD study group. Cardiovascular disease risk factors in HIV patients--association with antiretroviral therapy. Results from the DAD study. AIDS. 2003 May 23;17(8):1179-93. doi: 10.1097/01.aids.0000060358.78202.c1. PMID 12819520
- [Result] Chene G, Sterne JA, May M, Costagliola D, Ledergerber B, Phillips AN, Dabis F, Lundgren J, D'Arminio Monforte A, de Wolf F, Hogg R, Reiss P, Justice A, Leport C, Staszewski S, Gill J, Fatkenheuer G, Egger ME; Antiretroviral Therapy Cohort Collaboration. Prognostic importance of initial response in HIV-1 infected patients starting potent antiretroviral therapy: analysis of prospective studies. Lancet. 2003 Aug 30;362(9385):679-86. doi: 10.1016/s0140-6736(03)14229-8. PMID 12957089
- [Result] Friis-Moller N, Sabin CA, Weber R, d'Arminio Monforte A, El-Sadr WM, Reiss P, Thiebaut R, Morfeldt L, De Wit S, Pradier C, Calvo G, Law MG, Kirk O, Phillips AN, Lundgren JD; Data Collection on Adverse Events of Anti-HIV Drugs (DAD) Study Group. Combination antiretroviral therapy and the risk of myocardial infarction. N Engl J Med. 2003 Nov 20;349(21):1993-2003. doi: 10.1056/NEJMoa030218. PMID 14627784
- [Result] Miller V, Phillips AN, Clotet B, Mocroft A, Ledergerber B, Kirk O, Ormaasen V, Gargalianos-Kakolyris P, Vella S, Lundgren JD. Association of virus load, CD4 cell count, and treatment with clinical progression in human immunodeficiency virus-infected patients with very low CD4 cell counts. J Infect Dis. 2002 Jul 15;186(2):189-97. doi: 10.1086/341466. Epub 2002 Jul 3. PMID 12134254
- [Result] Egger M, May M, Chene G, Phillips AN, Ledergerber B, Dabis F, Costagliola D, D'Arminio Monforte A, de Wolf F, Reiss P, Lundgren JD, Justice AC, Staszewski S, Leport C, Hogg RS, Sabin CA, Gill MJ, Salzberger B, Sterne JA; ART Cohort Collaboration. Prognosis of HIV-1-infected patients starting highly active antiretroviral therapy: a collaborative analysis of prospective studies. Lancet. 2002 Jul 13;360(9327):119-29. doi: 10.1016/s0140-6736(02)09411-4. PMID 12126821
- [Result] Ledergerber B, Mocroft A, Reiss P, Furrer H, Kirk O, Bickel M, Uberti-Foppa C, Pradier C, D'Arminio Monforte A, Schneider MM, Lundgren JD; Eight European Study Groups. Discontinuation of secondary prophylaxis against Pneumocystis carinii pneumonia in patients with HIV infection who have a response to antiretroviral therapy. Eight European Study Groups. N Engl J Med. 2001 Jan 18;344(3):168-74. doi: 10.1056/NEJM200101183440302. PMID 11188837
- [Derived] Mocroft A, Geressu A, Beguelin C, Llibre JM, Lazarus JV, Tomazic J, Smidt J, Parczewski M, Brannstrom J, Sedlacek D, Degen O, van der Valk M, Paduta D, Flamholc L, Schmid P, Orkin C, Nielsen LN, Hoffmann C, Beniowski M, Oprea C, Begovac J, Peters L. The role of HIV/hepatitis B virus/hepatitis C virus RNA+ triple infection in end-stage liver disease and all-cause mortality in Europe. AIDS. 2023 Jan 1;37(1):91-103. doi: 10.1097/QAD.0000000000003406. Epub 2022 Oct 18. PMID 36476454
- See also: EuroSIDA — http://www.chip.dk/EuroSIDA